# Statistical Analysis Plan

## 209141

Phase II randomized, observer-blind, placebo-controlled, multi-country study in healthy non-pregnant women 18-45 years of age to evaluate the safety, reactogenicity and immunogenicity of a 1st intramuscular dose of GSK Biologicals' investigational RSV maternal vaccine (GSK388550A) when given alone and given in co-administration with a single intramuscular dose of Boostrix (US formulation SB776423 or ex-US formulation SB263855) and to evaluate the safety, reactogenicity and immunogenicity of a 2nd dose of the RSV maternal vaccine.

**EudraCT number:** 2019-002258-22

**Date of Document:** 03 DECEMBER 2020

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| | Statistical Analysis Plan Amendment 4 |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | Phase II randomized, observer-blind, placebo-controlled, multi-country study in healthy non-pregnant women 18-45 years of age to evaluate the safety, reactogenicity and immunogenicity of a 1st intramuscular dose of GSK Biologicals' investigational RSV maternal vaccine (GSK388550A) when given alone and given in co-administration with a single intramuscular dose of Boostrix (US formulation SB776423 or ex-US formulation SB263855) and to evaluate the safety, reactogenicity and immunogenicity of a 2nd dose of the RSV maternal vaccine. |
| eTrack study number and<br>Abbreviated Title | 209141 (RSV MAT-011) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 21 October 2019 |
| Date of Statistical Analysis plan amendment | Amendment 2 Final: 28 February 2020 |
| | Amendment 3 Final: 03 April 2020 |
| | Amendment 4 Final: 03 December 2020 |
| APP 9000058193 | Statistical Analysis Plan Template V4 (Effective date: 3June2019) |

# 209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# **TABLE OF CONTENTS**

| | | | | | | | PAGE |
|---|---|---|---|---|---|---|---|
| LIS | T OF A | ABBREVI | ATIONS | | | | 6 |
| 1. | DOC | JMENT H | ISTORY | | | | 9 |
| 2. | OBJE | CTIVES/ | ENDPOINTS | <b></b> | | | 9 |
| 3. | STUE | Y DESIG | N | | | | 11 |
| 4. | ΔΝΔΙ | VSIS SE | TS (AMENID) | FD 03-DFC | :-2020) | | 15 |
| Τ. | 4.1. | | | | | | |
| | | 4.1.1. | | | | | |
| | | 4.1.2. | | | Set | | |
| | 4.2. | | | | n Analysis Sets | | |
| | | 4.2.1. | | | sed Set (ES) | | |
| | | 4.2.2. | Flimination | from Per-r | protocol analysis Se | t (PPS) | 16 |
| | | | 4.2.2.1. | | subjects from Per-pr | | |
| | | | | | | | 16 |
| | | 4.2.3. | Elimination | | ted safety set | | |
| | | | 4.2.3.1. | | subjects | | |
| | | | | | Solicited safety se | | |
| 5. | | | | | | | |
| | 5.1. Demography | | | | | | |
| | | 5.1.1. | | | | | |
| | | 5.1.2. | | | ons | | |
| | 5.2. | | | | | | 19 |
| | | 5.2.1. | Analysis of | fimmunoge | enicity planned in the | e protocol | |
| | | | | | 020) | | |
| | | 5.2.2. | | | ons | | |
| | | | 5.2.2.1. | | roup analysis | | |
| | | | 5.2.2.2. | | e difference betwee | | |
| | 5.3. | | | | nicity | | 22 |
| | | 5.3.1. | Analysis of | r safety and | reactogenicity plan | ined in the | 00 |
| | | <b>5</b> 00 | | | B-DEC-2020) | | |
| | | 5.3.2. | | | ons | | |
| | | | 5.3.2.1. | | solicited events | | |
| | | | 5.3.2.2. | | Unsolicited Advers | | 25 |
| | | | 5.3.2.3. | | Solicited and Unsol | | 0.5 |
| | | | F 2 2 4 | | | | |
| | | | 5.3.2.4. | Other anal | ysis | | 26 |
| 6. | ANAL | YSIS INT | ERPRETAT | ION | | | 26 |
| 7. | CONI | DUCT OF | ANALYSES | | | | 26 |
| • | 7.1. | | | | | | |
| | | 7.1.1. | | | | | |
| | 7.2. | | al considera | tions for int | erim analyses | | 27 |

# 209141 (RSV MAT-011)

| 8. | CHAN | IGES FRO | M PLANNE | ED ANALYSES (AMENDED 03-DEC-2020) | 27 |
|---|---|---|---|---|---|
| 9. | | | | ERIVATION RULES AND STATISTICAL | 00 |
| | 9.1. | | | | |
| | | 9.1.1. | | enicity (Amended 03-DEC-2020) | 20 |
| | | 9.1.1.1. | | assays cut-offs for humoral immunity (Antibody | 20 |
| | 9.2. | Statistica | | tion) (Amended 03-DEC-2020) | |
| 10 | ∧ NINI⊏ | VEC | | | 20 |
| 10. | 10.1. | | | tandard data derivations and statistical methods | |
| | 10.1. | | | events to vaccine doses | |
| | | 10.1.1. | | of missing data | |
| | | 10.1.2. | | Dates | |
| | | | | Laboratory data | |
| | | | 10.1.2.2. | Solicited adverse events (Amended 03-DEC- | 32 |
| | | | 10.1.2.3. | 2020) | 32 |
| | | | 10.1.2.4. | Unsolicited adverse events | 32 |
| | | 10.1.3. | | ation | |
| | | 10.1.5. | 10.1.3.1. | Age at vaccination in years | |
| | | | 10.1.3.1. | Weight | |
| | | | 10.1.3.2. | Height | |
| | | | 10.1.3.4. | Body mass index (BMI) | |
| | | | 10.1.3.4. | Temperature | |
| | | | 10.1.3.6. | Numerical serology results | |
| | | | 10.1.3.0. | Geometric mean titres (GMTs) and | 54 |
| | | | 10.1.5.7. | concentrations (GMCs) | 34 |
| | | | 10.1.3.8. | Onset day | |
| | | | 10.1.3.9. | | |
| | | | | Counting rules for combining solicited and | 04 |
| | | | 10.1.0.10. | unsolicited adverse events | 34 |
| | | | 10 1 3 11 | Counting rules for occurrences of solicited | |
| | | | 10.1.0.11. | adverse events | 35 |
| | | 10.1.4. | Display of | decimals | |
| | | | 10.1.4.1. | Percentages | |
| | | | 10.1.4.2. | Differences in percentages | |
| | | | 10.1.4.4. | Serological summary statistics | |
| | | 10.1.5. | | methodology | |
| | | | | Exact confidence intervals around proportions | |
| | | | | Standardized asymptotic confidence intervals | |
| | | | | around differences in proportions | 37 |
| | 10.2. | TFL TOO | <b>)</b> | | |
| 11 | RFFF | RENCES | | | 38 |

# 209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study objectives and endpoints (Amended 03-DEC-2020) | 9 |
| Table 2 | Study groups, pooled study groups (Amended 03-DEC-2020) | 13 |
| Table 3 | Study groups, treatment and epochs foreseen in the study (Amended 03-DEC-2020) | 14 |
| Table 4 | Elimination code and condition (Amended 03-DEC-2020) | 16 |
| Table 5 | Intensity scales for solicited symptoms in adults | 24 |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# **LIST OF FIGURES**

| | PAGE |
|---------------------------------------------------|------|
| ire 1 Study design overview (Amended 03-DEC-2020) | 11 |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# **LIST OF ABBREVIATIONS**

**Ab** Antibody

**AE(s)** Adverse Event(s)

**AE** Adverse Event

**Anti-** Antibodies against

**BS H** Blood Sample Humoral

**CDC** Centers for Disease Control

CI Confidence Interval

CLS Clinical Laboratory Sciences

**CoP** Correlate of Protection

**D** Diphtheria

dTpa Diphtheria, Tetanus and acellular Pertussis

**eCRF** electronic Case Report Form

**ELISA** Enzyme-Linked Immunosorbent Assay

**EoS** End of Study

eTDF Electronic Temperature excursion Decision Form

**Ex-US** Outside the US

**FDA** Food and Drug Administration, United States of America

**FHA** Filamentous Hemagglutinin

FU Follow-up

GCP Good Clinical Practice

GMC Geometric Mean Concentration

**GMT** Geometric Mean Titer

**GSK** GlaxoSmithKline

IAF Informed Assent Form

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

**IB** Investigator Brochure

**ICF** Informed Consent Form

**ICH:** International Council on Harmonisation

**IEC** Independent Ethics Committee

IgG Immunoglobulin

IM Intramuscular

IMP Investigational Medicinal Product

IND Investigational New Drug

**IRB** Institutional Review Board

LAR Legally Acceptable Representative

**LSLV** Last Subject Last Visit

MACDP Metropolitan Atlanta Congenital Defects Program

**MedDRA** Medical Dictionary for Regulatory Activities

**Nab** Neutralizing antibody

**PCD** Primary Completion Date

**PP** Per protocol

**PRN** Pertactin

**PRO** Patient Related Outcomes

PT Pertussis Toxoid

**RRA** Recruitment/Randomisation Agreement

**RSV** Respiratory Syncytial Virus

**RSVPreF3** RSV maternal vaccine

**SAE:** Serious Adverse Event

**SBIR** Source data Base for Internet Randomisation

**SD** Standard Deviation

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

**SDV** Source Document Verification

**SmPC** Summary of Product Characteristics

**SPM** Study Procedures Manual

**SRT** Safety Review Team

T Tetanus

**UP** Urine Pregnancy Test

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|--------------------------|
| 03 DEC 2020 | Amendment 4 | Amendment 4: 30-AUG-2020 |
| 03 APR 2020 | Amendment 3 | Amendment 3: 03-APR-2020 |
| 28 FEB 2020 | Amendment 2 | Amendment 2: 28-FEB-2020 |
| 21 OCT 2019 | first version | Final: 28 JUN 2019 |

# 2. OBJECTIVES/ENDPOINTS

# Table 1 Study objectives and endpoints (Amended 03-DEC-2020)

| Obje | ectives | Endpoints |
|---|---|---|
| Prim | nary (US + ex-US data to be pooled) | |
| Safe | ety | Safety |
| • | To evaluate the safety and reactogenicity of 2 dose levels (60 and 120 μg) of RSVPreF3 when given alone or co-administered with dTpa from Vaccination up to Day 31. | Occurrence of any Adverse Events (AEs) from Vaccination to Day 31: Occurrence of each solicited local AEs at the site of injection in both limbs from Vaccination to Day 8; Occurrence of solicited general AEs from Vaccination to Day 8; Occurrence of any unsolicited AEs from Vaccination to Day 31; Occurrence of Serious Adverse Events (SAEs) from Vaccination to Day 31. |
| • | To evaluate the safety of a 2 <sup>nd</sup> dose of RSVPreF3 given from 12 up to18 months post 1st Dose up to Day 31 days post 2 <sup>nd</sup> dose vaccination | <ul> <li>Occurrence of any AEs from 2<sup>nd</sup> dose to Day 31 post-2<sup>nd</sup> dose vaccination, for all subjects:</li> <li>Occurrence of each solicited local AE at the site of injection in both deltoids from 2<sup>nd</sup> dose vaccination to Day 8 post-2<sup>nd</sup> dose vaccination</li> <li>Occurrence of solicited general AEs from 2<sup>nd</sup> dose vaccination to Day 8 post 2<sup>nd</sup> dose vaccination</li> <li>Occurrence of any unsolicited AEs from 2<sup>nd</sup> dose to Day 31 post-2<sup>nd</sup> dose vaccination</li> <li>Occurrence of Serious Adverse Events (SAEs) from 2<sup>nd</sup> dose vaccination to Day 31 post 2<sup>nd</sup> dose vaccination.</li> </ul> |
| lmm | unogenicity | Immunogenicity |
| • | To evaluate the humoral immune response to 2 dose levels (60 and 120 µg) of RSVPreF3 when given alone and co-administered with dTpa, at Screening, Day 8 and Day 31 post 1st dose vaccination | <ul> <li>RSV A neutralizing antibody titers at Screening,<br/>Day 8 and Day 31 in all groups</li> <li>RSV IgG antibody concentrations at Screening, Day 8 and Day 31.</li> </ul> |
| _ | ondary (US and ex-US data to be considered pooled, | 1 |
| Safe | ty | Safety |
| • | To evaluate the safety and reactogenicity of 2 dose levels (60 and 120 μg) of RSVPreF3 when given | Occurrence of any AEs from Vaccination to Day 31, for all subjects: |

# 209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| Objectives | Endpoints |
|---|---|
| alone or co-administered with dTpa from 1st dose vaccination up to Day 31 by formulation. | Occurrence of each solicited local AE at the site of injection in both limbs from Vaccination to Day 8 |
| | Occurrence of solicited general AEs from<br>Vaccination to Day 8 |
| | Occurrence of any unsolicited AEs from<br>Vaccination to Day 31 |
| | <ul> <li>Occurrence of Serious Adverse Events (SAEs) from<br/>Vaccination to Day 31.</li> </ul> |
| <ul> <li>To evaluate the safety of 2 dose levels (60 and<br/>120 µg) of RSVPreF3 when given alone and co-<br/>administered with dTpa compared to dTpa-Placebo<br/>groups from 1st dose vaccination up to Day 181.</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |
| <ul> <li>To evaluate the safety of 2 dose levels (60 and<br/>120 µg) of RSVPreF3 when given alone and co-<br/>administered from Vaccination up to Day 181 by<br/>formulation.</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |
| <ul> <li>To evaluate the safety of RSVPreF3 (pooled for all<br/>groups receiving RSVPreF3) for the 1<sup>st</sup> dose<br/>vaccination.</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |
| To evaluate the safety of 2 <sup>nd</sup> dose of RSVPreF3 given from 12 to up to 18 months post 1 <sup>st</sup> dose vaccination up to Day 181 post 2 <sup>nd</sup> dose vaccination. | Occurrence of SAEs from 2 <sup>nd</sup> dose vaccination up to Day 181 post-2 <sup>nd</sup> dose vaccination. |
| Immunogenicity | Immunogenicity |
| <ul> <li>To evaluate the humoral immune response and<br/>persistence to 2 dose levels (60 and 120 μg) of<br/>RSVPreF3 when given alone and co-administered<br/>with dTpa at Screening, Day 8, and Day 31 post 1st<br/>dose vaccination, and at 12 to 18 months by<br/>formulation.</li> </ul> | <ul> <li>RSV A neutralizing antibody titers at Screening, Day 8, Day 31, and a single timepoint between 12 to 18 months post 1st vaccination.</li> <li>RSV IgG antibody concentrations at Screening, Day 8, Day 31, and a single timepoint between 12 to 18 months post 1st vaccination.</li> </ul> |
| <ul> <li>To evaluate the humoral immune response to the<br/>pertussis component of the dTpa vaccine when<br/>given alone and co-administered with 2 dose levels<br/>(60 and 120 µg) of RSVPreF3 at Screening and Day<br/>31 post 1st dose vaccination by formulation.</li> </ul> | Antibody concentrations against pertussis toxoid<br>(anti-PT), filamentous hemagglutinin (anti-FHA), and<br>pertactin (anti-PRN) concentrations at Screening<br>and Day 31. |
| <ul> <li>To evaluate the humoral immune response to the<br/>diphtheria (D) component of dTpa vaccine when<br/>given alone and co-administered with 2 dose levels<br/>(60 and 120 µg) of RSVPreF3 at Screening and Day<br/>31 post 1st dose vaccination by formulation.</li> </ul> | Anti-D concentrations at Screening and Day 31. |
| <ul> <li>To evaluate the humoral immune response to the<br/>tetanus (T) component of dTpa vaccine when given<br/>alone and co-administered with 2 dose levels (60<br/>and 120 μg) of RSVPreF3 at Screening and Day 31<br/>post 1st dose vaccination by formulation.</li> </ul> | Anti-T concentrations at Screening and Day 31. |
| <ul> <li>To evaluate the humoral immune response of a 2<sup>nd</sup> dose vaccination of RSVPreF3 (120 μg), following a first dose vaccination of either 60 μg or 120 μg.</li> </ul> | <ul> <li>RSV A neutralizing antibody titers concentrations 31 days post 2<sup>nd</sup> dose vaccination.</li> <li>RSV IgG antibody concentrations 31 days post 2<sup>nd</sup> dose vaccination.</li> </ul> |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| Objectives | Endpoints |
|---|---|
| Tertiary | |
| If necessary, additional testing to further characterize the be performed. | response to the RSV maternal investigational vaccine will |

# 3. STUDY DESIGN

Figure 1 Study design overview (Amended 03-DEC-2020)



Note: study groups labeled X = ex-US; study groups labeled U = US. V = visit, C = phone contact

>= Vaccination; N = number of subjects; V = Visit; D = Day; AE = adverse event; UP = Urine pregnancy test; CHS = Chemical/Hematological Screening, FU = follow-up

BSH = blood sample (5 mL) for humoral immune responses (RSV-A neutralization and RSV IgG antibody concentrations at Screening, Visit 2, [Day 8] Visit 3, [Day 31], Visit 4, [up to D7 prior to 2<sup>nd</sup> vaccination], and Visit 6 [D31 post 2<sup>nd</sup> vaccination]

dTpa ELISAs at Screening and Visit 3 [Day 31])

- \* All subject groups will be given RSV 120mcg and subjects will be followed in an open labeled study
- \*\* Hematological and biochemical laboratory testing at Visit 4 (D -7 up to and including 2<sup>nd</sup> dose vaccination) at the investigator's discretion

The study will be conducted with 2 formulations of dTpa, dTpa\_300 (in the US) and dTpa\_500 (ex-US) [Christy, 1995].

<sup>\*\*\*</sup>There will be no follow-up between C1 and V4. New medical history and relevant new safety events during this period will be recorded at visit 4 for subjects who agree to the study extension and sign the informed consent addendum.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

Approximately 500 eligible subjects (250 in the US and 250 ex-US) will be enrolled. Of these, approximately 250 subjects will be randomized to 5 US study groups in a 1:1:1:1:1 ratio using SBIR, and the remaining approximately 250 will be randomized to 5 ex-US study groups in a 1:1:1:1:1 ratio using SBIR. The randomization algorithm will use a minimization procedure by treating study formulation (US and ex-US) as a stratification factor, and age at the time of vaccination (18-32 or 33-45 years of age) and center as minimization factors

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the schedule of activities, are essential and required for study conduct.

- Type of study: self-contained
- Experimental design:
  - Primary Vaccination: multi-centric study, multi-country Phase II, observer-blind, randomized, with 5 parallel groups in each formulation (US, ex-US).

Study Extension: multi-centric study, multi-country Phase II, open label, with all 5 parallel groups in each formulation (US, ex-US) receiving the experimental RSV maternal (120µg) vaccine.

- Duration of the study: The primary study will be approximately 6 months for each enrolled subject, the duration of the study extension will be 18 up to 24 months.
  - Primary Vaccination
    - Epoch 001: Screening
    - Epoch 002: Primary vaccination starting at Visit 1 (Day 1) and ending just before the Visit 3 (Day 31)
    - Epoch 003: Follow-up after Visit 3 (Day 31) to Phone Contact 1 on (Day 181)
  - End of Primary Study: Subjects must sign the ICF addendum to join the study extension.
  - Study Extension: 6-month period starting at the beginning of 12 months up to the beginning of 18<sup>th</sup> month after Visit 1 (≥12 to <18 months)</li>
    - Epoch 004: 2nd dose vaccination starting from Visit 4 (up -7 days prior to vaccination) to Visit 6 (Day 31 post 2nd dose vaccination)
    - Epoch 005: 2nd dose vaccination Study Follow-up 2 starting after Visit 6 (Day 31 post 2nd dose vaccination) and ending at Phone Contact 3 (Day 181 post 2nd vaccination).
- Primary completion Date (PCD): Visit 3 (Day 31) or last visit of Primary Epoch 002 Refer to list of abbreviations for the definition of PCD.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

• End of Study (EoS): Last testing results released of samples collected at Visit 6, to occur no later than 8 months after last subject last visit (LSLV), which occurs with phone contact 3 on Day 181 post 2<sup>nd</sup> vaccination.

Refer to list of abbreviations for the definition of EoS.

# • Study groups:

Table 2 Study groups, pooled study groups (Amended 03-DEC-2020)

| Pooled Groups<br>label in tables | Pooled definition for footnote | Group label in tables | Group definition for footnote |
|---|---|---|---|
| RSV120_dTpa | Subjects who received | XRSV120_dTpa | Subject who received RSV MAT 120 and<br>Boostrix-ex-US (dTpa_500) |
| K3V120_U1pa | RSV120 and dTpa | URSV120_dTpa | Subjects who received RSV MAT 120 and<br>Boostrix-US (dTpa_300) |
| RSV120_Placebo | Subjects who received | XPlacebo_RSV120 | Subject who received RSV MAT 120 and Placebo |
| 1.5V 12U_F lacebo | RSV120 and placebo | UPlacebo_RSV120 | Subject who received RSV MAT 120 and Placebo |
| RSV60_ dTpa | Subjects who received | XRSV60_dTpa | Subjects who received RSV MAT 60 and<br>Boostrix-ex-US (dTpa_500) |
| 113700_ u i pa | RSV60 and dTpa | URSV60_dTpa | Subjects who received RSV MAT 60 and<br>Boostrix-US (dTpa_300) |
| RSV60_Placebo | Subjects who received | XPlacebo_RSV60 | Subjects who received RSV MAT 60 and Placebo |
| TOVOO_I lacebo | RSV60 and placebo | UPlacebo_RSV60 | Subject who received RSV MAT 60 and Placebo |
| dTpa_Placebo | Subjects who received | XPlacebo_dTpa | Subject who received <i>Boostrix</i> -ex-US (dTpa_500) and Placebo |
| итра_гіасеро | Boostrix(dTpa) and<br>Placebo | UPlacebo_dTpa | Subject who received <i>Boostrix</i> -US (dTpa_300) and Placebo |
| RSV_placebo | Subjects who received<br>RSV60 and placebo<br>combined with subjects who<br>received RSV120 and<br>placebo | | |
| RSV_dTpa | Subjects who received<br>RSV60 and dTpa combined<br>with subjects who received<br>RSV 120 and dTpa | | |

Table 3 Study groups, treatment and epochs foreseen in the study (Amended 03-DEC-2020)

| | | | | Treatment name 2 | Epochs<br>(Blinding) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Groups | Number of subjects | Age<br>(Min-<br>Max) | Treatment name 1 | | Epoch 001<br>(Screening) | Epoch 002<br>(observer-<br>blind) | Epoch 003<br>(single-<br>blind) | Epoch<br>004 (open<br>Label) | Epoch 00<br>5<br>(open<br>study) |
| XRSV120_dTpa | 50 | 18 – 45<br>years | RSV MAT 120<br>Boostrix-ex-US<br>(dTpa_500) | RSV MAT 120 | х | х | х | Х | х |
| Xplacebo_RSV120 | 50 | 18 – 45<br>years | RSV MAT 120<br>Placebo | RSV MAT 120 | х | х | х | Х | Х |
| XRSV60_dTpa | 50 | 18 – 45<br>years | RSV MAT 60<br>Boostrix-ex-US<br>(dTpa_500) | RSV MAT 120 | х | х | х | х | Х |
| Xplacebo_RSV60 | 50 | 18 – 45<br>years | RSV MAT 60<br>Placebo | RSV MAT 120 | х | х | х | Х | Х |
| Xplacebo_dTpa | 50 | 18 – 45<br>years | Boostrix-ex-US<br>(dTpa_500)<br>Placebo | RSV MAT 120 | х | х | х | х | х |
| URSV120_dTpa | 50 | 18 – 45<br>years | RSV MAT 120<br>Boostrix-US<br>(dTpa_300) | RSV MAT 120 | х | х | х | х | х |
| Uplacebo_RSV120 | 50 | 18 – 45<br>years | RSV MAT 120<br>Placebo | RSV MAT 120 | х | х | х | Х | Х |
| URSV60_dTpa | 50 | 18 – 45<br>years | RSV MAT 60<br>Boostrix-US | RSV MAT 120 | х | х | х | Х | Х |
| Uplacebo_RSV60 | 50 | 18 – 45<br>years | RSV MAT 60<br>Placebo | RSV MAT 120 | х | х | х | Х | Х |
| Uplacebo_dTpa | 50 | 18 – 45<br>years | Boostrix-US<br>(dTpa_300)<br>Placebo | RSV MAT 120 | x | х | х | Х | Х |

3 December 2020 14

- **Control:** (active comparator).
- **Treatment allocation**: (randomised stratified).
- **Blinding:** As described in Table 3.
- **Data collection**: standardised Electronic Case Report Form (eCRF). Solicited symptoms will be collected using a subject paper Diary (pDiary).
- Safety monitoring:

If the investigator becomes aware of a holding rule being met, he/she will suspend vaccination and will inform GSK immediately.

# 4. ANALYSIS SETS (Amended 03-DEC-2020)

## 4.1. Definition

For purposes of analysis, the following analysis sets are defined:

| Analysis Set | Description |
|---|---|
| Enrolled | Subjects who agreed to participate in a clinical study after completion of the |
| Emonod | informed consent process. And subject is not a screen failure. |
| Exposed | All subjects who received at least 1 dose of the study treatment. The allocation |
| Lxposed | in a group is done in function of the administered treatment. |
| | All subjects who received at least 1 dose of the study treatment to which they |
| Per Protocol | are randomised and have post-vaccination data minus subjects with protocol |
| | deviations that lead to exclusion |
| Solicited Safety | All subjects who received at least 1 dose of the study treatment (Exposed Set) |
| Solicited Salety | who have solicited safety data |

## 4.1.1. Exposed Set

The ES will include all subjects who received at least 1 dose of the study treatment.

• A **safety** analysis based on the ES will include all subjects who received at least 1 dose of the study treatment.

# 4.1.2. Per Protocol Analysis Set

Per protocol analysis set will be defined by time points. It will include all subjects who received at least 1 dose of the study treatment to which they are randomised and have post-vaccination data minus subjects with protocol deviations that lead to exclusion at Screening, Day 8 and Day 31 post 1<sup>st</sup> dose, Visit 4 and Visit 6 post 2<sup>nd</sup> dose.

• An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available, if, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

Code 1030 (Study vaccine not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from PPS

# 4.2.2.1. Excluded subjects from Per-protocol analysis set

A subject will be excluded from the PPS analysis under the following conditions

Table 4 Elimination code and condition (Amended 03-DEC-2020)

| Code | Condition under which the code is used | Visit (timepoints)<br>where the code is<br>applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 800 | Fraudulent data | All | All |
| 900 | Invalid informed consent | All | All |
| 1030 | Study vaccine not administered at all | All | Safety, immunogenicity |
| 1040.Vx+* | Administration of concomitant vaccine(s) forbidden in the protocol | All | Immunogenicity |
| 1050 | Randomisation failure | All | Immunogenicity |
| 1060 | Randomisation code was broken | All | Immunogenicity |
| 1070** | Subjects got vaccinated with the correct vaccine but containing an incorrect volume | All | Immunogenicity |
| 1070** | Vaccination not according to protocol (site of injection, route of administration, wrong replacement of study treatment administered) | All | Immunogenicity |
| 1070** | Study treatment not prepared as per protocol (e.g. reconstitution) | All | Immunogenicity |
| 1070** | Other deviations related to wrong study treatment/administration/dose | eviations related to wrong study | |
| 1070** | Study treatment administered while All Immunogenicity contraindication | | Immunogenicity |
| 1080 | Vaccine temperature deviation | All | Immunogenicity |
| 1090 | | | Immunogenicity |
| 2010 | Protocol violation (inclusion/exclusion criteria) DOB – VAC – 18-45 years | All | Immunogenicity |

# 209141 (RSV MAT-011)

# Statistical Analysis Plan Amendment 4

| Code | Condition under which the code is used | Visit (timepoints)<br>where the code is<br>applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 2150 | Failure to report safety events per protocol | All | Safety |
| 2040.Vx+* | Administration of any medication forbidden by the protocol | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |
| 2040.Vx+* | Device, excluded by the protocol, was administered | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 6 | Immunogenicity |
| 2050.Vx+* | Intercurrent medical conditions which are exclusionary as per protocol | Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |
| 2060.Vx+* | Concomitant infection related to the vaccine which may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 6 | Immunogenicity |
| 2070.Vx+* | Concomitant infection not related to the vaccine but may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |
| 2090.Vx | Subjects did not comply with blood sample schedule: • For PPS at Day 8, check the interval from vaccination to day 8 BS = 7 - 10 days; • For PPS at Day 31, check the interval from vaccination to day 31 BS = 30 - 45 days; • For PPS at Visit 6, check the interval from Visit to Visit 5 • BS = 365 - 548 days; | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |
| 2100.Vx | Serological results not available post-<br>vaccination | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |
| 2120.Vx* | Obvious incoherence or abnormality or error in data Visit 2/Day 8 Visit 3/Day 31 Visit 4 Visit 6 | | Immunogenicity |
| 2130.Vx | Testing performed on samples not aligned with ICF | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4<br>Visit 6 | Immunogenicity |

<sup>\*</sup>Attribution of these elimination codes to subject need CRDL review of individual listing

DOB-Date of Birth, VAC-Vaccination, BS- Blood Sample

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation Vx+ indicates subjects whose immunogenicity data will be eliminated from a specific visit onwards; Vx indicates subjects whose immunogenicity data will be eliminated from a specific visit.

#### 4.2.3. Elimination from solicited safety set

#### 4.2.3.1. **Excluded subjects**

## 4.2.3.1.1. Solicited safety set

Code 1030 (Study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used for identifying subjects eliminated from the solicited safety set.

#### 5. STATISTICAL ANALYSES

#### 5.1. **Demography**

### 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

These analyses will be performed on the Exposed set and on the Per protocol set for immunogenicity.

For all subjects, demographic characteristics (e.g., age at vaccination (18-32: 33-45 years), race and ethnicity, vaccination history will be summarized by overall and vaccine group using descriptive statistics.

- Frequency tables will be generated for categorical variables such as age
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height, weight and body mass index (BMI).

#### 5.1.2. Additional considerations

Demographic characteristics will also be summarized on Enrolled Set for web public disclosure.

Subject disposition will be summarized by group using descriptive statistics:

Number of subjects screened, randomised, vaccinated and withdrawn including withdrawal reasons in each group and overall will be tabulated.

Vital signs will be summarized by group using descriptive statistics at all timepoint(s) the information is collected on Exposed Set and Per-protocol Set.

Summary of important protocol deviations leading to elimination will be tabulated by group. An individual listing will also be provided.

Summary of medical history will be performed on Exposed Set by Medical Dictionary for Regulatory Activities (MedDRA) and preferred term.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

Summary of vaccination history will be performed on Exposed Set by using GSKDRUG dictionary.

Additional analyses by country and/or by site may be performed if deemed necessary

# 5.2. Immunogenicity

# 5.2.1. Analysis of immunogenicity planned in the protocol (*Amended 03-DEC-2020*)

The primary analysis on immunogenicity will be based on the Per Protocol set. If, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more, a second analysis based on the Exposed Analysis Set will be performed to complement the Per Protocol analysis.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled for the first vaccination) |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically pooled.</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI pooled.</li> </ul> |
| | <ul> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> </ul> |
| | The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentrations may be calculated at Screening, and/or Day 8, and/or Day 31 post 1st vaccination pooled for all subjects. |
| | A further exploratory between-groups analysis will be performed at Day 8 or Day 31 using an ANCOVA model by including study groups, study formulation (US and ex-US), age category, and level of antibodies at Screening as covariates. |
| Secondary | (US and ex-US data to be considered pooled, then separately for the first vaccination) |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically by formulation (US and ex-US) Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI by formulation (US and ex-US).</li> <li>Antibody titer/concentration will be displayed using reverse cumulative curves by</li> </ul> |
| | <ul> <li>formulation (US and ex-US).</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points by formulation (US and ex-US).</li> <li>Booster response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by group for each formulation (US and ex-US).</li> </ul> |
| | For the data collected for the second vaccination, the humoral immune response of RSV PreF3 will be summarized based on 2 dose level (60 and 120 µg) from the first vaccination. |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| Endpoint | Statistical Analysis Methods |
|---|---|
| | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically for prior and<br/>post 2<sup>nd</sup> dose vaccination</li> </ul> |
| | <ul> <li>Geometric mean of ratios of antibody titer/concentrations at individual post- 2<sup>nd</sup> dose<br/>vaccination time point (visit 6) over prior 2<sup>nd</sup> dose vaccination time point (visit 4) will be<br/>tabulated with 95% CI</li> </ul> |
| | <ul> <li>Antibody titer/concentration will be displayed using reverse cumulative curves on prior and<br/>post 2<sup>nd</sup> vaccination</li> </ul> |
| | The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points including the visits from the first vaccination. |
| | Booster responses to PT, FHA and PRN antigens are defined as: |
| | <ul> <li>For subjects with pre-vaccination antibody concentration below the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the assay cut-offs,</li> </ul> |
| | <ul> <li>For subjects with pre-vaccination antibody concentration between the assay cut-offs and<br/>below 4 times the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the<br/>pre-vaccination antibody concentration, and</li> </ul> |
| | <ul> <li>For subjects with pre-vaccination antibody concentration ≥ 4 times the assay cut-offs:<br/>post-vaccination antibody concentration ≥2 times the pre-vaccination antibody<br/>concentration.</li> </ul> |
| | <ul> <li>The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for each formulation (US and ex-US).</li> </ul> |
| | <ul> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo<br/>in terms of anti-PT, anti-FHA, anti-PRN, anti-D, anti-T will be calculated at Screening<br/>and Day 31 pooled for all subjects and by formulation (US and ex-US).</li> </ul> |
| | <ul> <li>A further exploratory between-groups analysis will be performed at Day 31 using an<br/>ANCOVA model by including study groups, study formulation (US and ex-US), age<br/>category, and level of antibodies at Screening as covariates.</li> </ul> |
| | <ul> <li>For Boostrix booster response to antigens PT, FHA and PRN, the two-sided<br/>standardized asymptotic 95% CI for the group differences in the percentage of<br/>subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine<br/>group and (minus) the dTpa Placebo vaccine group on Day 31 post vaccination will<br/>be calculated for each formulation.</li> </ul> |
| | <ul> <li>For Boostrix seroprotection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for each formulation.</li> </ul> |
| Tertiary | Will be described in a Statistical Analysis Plan finalised before database unblinding/freezing. |

<sup>\*</sup>The statistical method will not be applied to primary endpoint. For detailed rationale, refer to Section 8.

\*\*pooled group definition is detailed in Table 2

## 5.2.2. Additional considerations

# 5.2.2.1. Between group analysis

The Non-inferiority on RSV-A neutralizing antibody titers at 31 days post 1<sup>st</sup> vaccination in the co-administration of RSVPreF3 vaccine + *Boostrix* compared to RSV+ Placebo will be evaluated based on the criterion below:

The criterion to evaluate non-inferiority with respect to RSV-A neutralizing antibody titers is that the upper limits of the 95% CI on the GMT ratio (RSVPreF3 +*Placebo* divided by RSVPre3 + Boostrix) is less than or equal to 1.5 at 31 days post vaccination.

Following model will be applied to RSVPreF3 IgG antibody concentrations and RSV-A neutralizing antibody titers.

For the analysis of subjects at visit 3 (Day 31), the model will be explored and fitted via the procedure according to the following code:

```
PROC glm data=sero;

CLASS group;

MODEL log_val = baseline group age_cat country_US country_BE

Output out= pred;

LSMEANS group/pdiff cl alpha=0.1;

RUN;
```

where **log\_val** represents the log-transformed antibody value of the immunogenicity variable at a given post baseline timepoint (Day 8) or (Day 31), **baseline** is prevaccination logarithm10 transformation of the concentrations/titers, **group** indicates the study group, pooled groups (US and ex-US) will considered in model then separate by formulation. **age\_cat** is indicator variable (0/1) and will be treated as continuous in the model, age\_cat equals 0 if the age category at vaccination between 18 - 32 years, otherwise age\_cat equals 1 if age category is between 33 - 45 years at vaccination. **Country\_US** is indicator variable (0/1) and will treated as continuous in the model, if subject from US, then variable will equal to 1, otherwise equals to 0, **Country\_BE** is indicator variable (0/1) and will treated as continuous in model, if subject from BE, then variable equals to 1, otherwise equals to 0, if subject is from Canada, above two indicators equal to 0. The inclusion of age category at vaccination, in the model depends on the availability of the variable and the necessity, therefore, the above SAS code serves as a reference and may be adjusted according to the analysis needs.

When considering group as separated by Boostrix formulation, remove Country\_US and Country\_BE from model.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

GMT/GMC ratios between vaccine groups obtained using above model will be calculated by exponentiating mean difference of logarithm- transformed titres. The 90% CI and 95% CI for GMT/GMC ratio will be obtained by exponential-transformation of the CI for the group least square mean of the log-transformed titres/concentration from the above model.

# 5.2.2.2. Percentage difference between two groups

The percentage difference of response rate in terms of antigen PT, FHA and PRN [Camargo, 1984; Melville, 1983], together with the two-sided standardized asymptotic 95% CI in the RSVPreF3 dTpa group (minus) the dTpa Placebo group on Day 31 will be provided.

The percentage difference of seroprotection rate in terms of antigen D and antigen T [Vidor, 2008] with the two-sided standardized asymptotic 95% CI for RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group by formulation at Day 31 will be calculated.

# 5.3. Analysis of safety and reactogenicity

# 5.3.1. Analysis of safety and reactogenicity planned in the protocol (*Amended 03-DEC-2020*)

The following safety analyses will be performed based on the Solicited Safety or Exposed Sets. The following safety analysis will be performed on the pooled data then the US and ex-US separately.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled) |
| | For each group with 1 <sup>st</sup> dose vaccination of RSVPreF3 (two dose levels) when given alone or co-ad with dTpa; the following points will be analysed for 1 <sup>st</sup> and 2 <sup>nd</sup> dose vaccination. |
| | The percentage of subjects with at least one local AE on left or right arm with at least one general AE and with any ("solicited or unsolicited") AE during the 7-day follow up period (the day of vaccination + 6 subsequent days) or 30 -day follow up period (the day of vaccination + 29 subsequent days) post 1st and 2nd vaccination period will be tabulated with exact 95% CI by study group. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits. |
| | The percentage of subjects reporting each individual solicited local AE (any grade, Grade 3 and those resulting in a medically attended visit) and solicited general AE (any grade, Grade 3, any related, Grade 3 related and those resulting in a medically attended visit) during the 7-day follow-up period (the day of vaccination + 6 subsequent days) will be tabulated based on maximum intensity for each group. |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (the day of vaccination + 6 subsequent days) will be tabulated for each group. Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| | Statistical Analysis Fight Amendment |
|---|---|
| Endpoint | Statistical Analysis Methods |
| | fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | The percentage of subjects with any unsolicited AEs during the 30-day follow-up period (the day of vaccination + 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) system organ classes (SOC) and preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit and leading to withdrawal from study. The verbatim term of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA SOC and Preferred Terms and reported during the 30-day follow-up period (the day of vaccination + 29 subsequent days) will be tabulated with exact 95% CI. SAEs will also be described in detail. |
| | The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period and during the 30-day follow-up period will be summarized by each group and pooled. |
| Secondary | (US and ex-US data to be considered pooled, then separately) |
| | For each group with 1 <sup>st</sup> dose vaccination of RSVPreF3 (two dose level) when given alone or coadministered with dTpa; the following points will be analysed for 1st and 2 <sup>nd</sup> dose vaccination. |
| | The percentage of subjects with at least one local AE with at least one general AE and with any ("solicited or unsolicited") AE during the 7-day or 30 -day follow-up as well any SAE up period to 180 days post 1st and 2nd vaccination time points will be tabulated with exact 95% CI by study group. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits and AEs leading to withdrawal from study. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA SOC and Preferred Terms and reported during the 30-day or 180-day follow-up period will be tabulated with exact 95% CI for each formulation (US and ex-US). |
| | The percentage of subjects reporting each individual solicited local AE on left or Right arms (any grade, Grade 3 and those resulting in a medically attended visit) and solicited general AE (any grade, Grade 3, any related, Grade 3 related and those resulting in a medically attended visit) during the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) will be tabulated based on maximum intensity for each group for each formulation (US and ex-US). |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period will be tabulated for each group for each formulation (US and ex-US). Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | For each formulation (US and ex-US), the percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e. on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) SOC and preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim term of unsolicited AEs will |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| Endpoint | Statistical Analysis Methods |
|---|---|
| | be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| Tertiary | Will be described in a Statistical Analysis Plan finalised before database unblinding/freezing. |

# 5.3.2. Additional considerations

# 5.3.2.1. Analysis of solicited events

The analysis of solicited events will be performed on Solicited Safety Set. The intensity of the following solicited events will be assessed as described:

Table 5 Intensity scales for solicited symptoms in adults

| Adults/Child (≥6 years) | | |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | collection questionna | ontained Clinical Outcome Assessment data aires or indices, which are protected by third and therefore have been excluded. |
| Redness at injection site | _ | |
| Swelling at injection site | _ | |
| Temperature* | _ | |
| Headache | | |
| Fatigue | | |
| Gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain) | | |

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

The maximum intensity of solicited administration site redness/swelling will be scored at GSK Biological as follows:

CCI - This section contained Clinical
Outcome Assessment data collection
questionnaires or indices, which are
protected by third party copyright laws and
therefore have been excluded.

Duration in days of solicited local and general adverse events within 7 days after vaccination will be tabulated by study group and overall, and if needed by age group. The derivation rule of duration in days for solicited events is detailed in section 10.1.3.9.

# 5.3.2.2. Analysis of Unsolicited Adverse Events

The analysis of unsolicited events will be performed on Exposed Set.

## 5.3.2.3. Combined Solicited and Unsolicited Adverse Events

The combined analysis of solicited and unsolicited events will be performed on Exposed Set. A summary of subjects with all combined solicited and unsolicited adverse events will be provided.

Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | Injection site pain | 10022086 |
| Redness | Injection site redness | 10022098 |
| Swelling | Injection site swelling | 10053425 |
| Fatigue | Fatigue | 10016256 |
| Fever | Fever | 10016558 |
| Headache | Headache | 10019211 |
| Gastrointestinal symptoms <sup>†</sup> | Gastrointestinal disorder | 10017944 |

Please note – to check for AE term in CDISC during dry run

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

<sup>†</sup>Gastrointestinal symptoms include nausea, vomiting, diarrhoea and/or abdominal pain.

# 5.3.2.4. Other analysis

Other safety analysis will be performed on Exposed Set.

Concomitant medications/products will be coded using the GSKDRUG dictionary. The number and percentage of subjects taking concomitant medications (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) within 7 days following vaccination, 30 days following vaccination and 12 months following vaccination will be summarized by group. A listing will also be provided.

## 6. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for most of these comparisons.

# 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

# 7.1.1. First and final study

Analyses to evaluate objectives and endpoints will be performed in steps.

- A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints pertaining to safety and immunogenicity up to Day 31 are available. At this point, the statistician will be unblinded (i.e. individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblind some specific subjects, the study will be considered as single-blind from this point onwards, subjects and investigators will be unblinded after Day 181 post 1st vaccination. The investigators will be provided with the individual data listings or with the randomization listings after Day 181.
- The **second analysis** will evaluate safety data and will be performed when **all subjects** have completed visits up to (and including) C1 (Day 181) and the data are available. From this point the study is unblinded and will continue as an open label study.
- The **third analysis** will evaluate safety and immunogenicity data and will be performed when **all subjects** have completed visits up to (and including) Visit 6 (Day 31 post 2<sup>nd</sup> dose vaccination) and the data are available. At this time, any available safety data will also be provided.
- The final end-of-study will be performed when all data for at least primary and secondary endpoints up to study conclusion at Day 181 post 2<sup>nd</sup> dose vaccination (C3) are available. An integrated clinical study report containing all available data will be written and made available to the investigators

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

The final study report will contain at least the final analyses of all primary and secondary endpoints. these analyses will be documented in in an amended study report. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed.

| Description | Disclosure Purpose (CTRS=public posting, SR=study report, internal) |
|---|---|
| First Analysis (E1_02) | Internal, Public disclosure |
| Second Analysis (E1_03) | Internal |
| Third Analysis (E1_04) | Internal |
| Final Analysis (E1 01) | Public disclosure, Study report |

# 7.2. Statistical considerations for interim analyses

NA

# 8. CHANGES FROM PLANNED ANALYSES (AMENDED 03-DEC-2020)

The calculation of GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3\_Placebo in terms of RSV-A Nab titers and RSV IgG antibody concentrations at Screening, Day 8 and Day 31 pooled for all subjects will be removed from analyses plan. We will report adjusted GMT/GMC ratio and their 95% CI which is generated from ANCOVA model.

Adjusted GMT/GMC ratio with both 90% CI and 95% CI which are generated from ANCOVA model will be reported in terms of RSV-A Nab titers and RSV IgG antibody concentrations.

The calculation of GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa\_Placebo groups in terms of antigens PT, FHA, PRN, D and T will be added at Day 31 pooled for all RSV formulation.

Lab assay cut-off of RSV-A Nab titers for humoral immunity will be reported by using both IU/ml (International units/millilitre) and ED60.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1

# 9.1. Data derivation

# 9.1.1. Immunogenicity (Amended 03-DEC-2020)

For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, analysis will exclude subjects with missing or non-evaluable measurements.

- For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude subjects with a missing or non-evaluable measurement.
- For the between group assessments, statistical model will be fitted based on the subjects having a result at both the baseline and the considered timepoint.

Following table shows all antigens will be analysed at considered time point for different treatment groups

| | Immunogenicity<br>Endpoints | Statistical Analysis Methods |
|---|---|---|
| | RSVPreF3 IgG antibody | (US and ex-US data to be considered pooled, then separately for the first vaccination, US and ex-US data to be pooled for second vaccination) |
| | concentration, and Neutralizing antibody titers against RSV-A | For the data collected for the second vaccination, the humoral immune response of RSV PreF3 will be summarized based on 2 dose levels (60 and 120 $\mu$ g) from the first vaccination. |
| RSVPreF3 | agamst NOV-A | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI</li> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> <li>A further exploratory between-groups of RSVPreF3 dTpa and BSV/RsF3 along in terms of RSVA A Neb titors and RSV/RsC antibody.</li> </ul> |
| | | RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentration, analysis will be performed at Day 8 and Day 31 post 1st dose using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates |

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

| | | Otatistical Analysis Flatt Amendment |
|---|---|---|
| | Immunogenicity<br>Endpoints | Statistical Analysis Methods |
| | Booster response to PT | For the subjects received RSVPreF3 dTpa and subjects received dTpa placebo |
| | <ul> <li>Booster response to FHA</li> <li>Booster response to PRN</li> </ul> | (US and ex-US data to be considered pooled, then separately for the first vaccination) |
| | | (US and ex-US data to be considered pooled for the second vaccination) |
| Boostrix<br>(dTpa) | | <ul> <li>Booster response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by group for US and ex-US pooled formulation and separately.</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-PT, anti-FHA, anti-PRN will be calculated between Day 31 post vaccination over Screening for US and ex-US pooled data and separately.</li> <li>For 1st vaccination, a further exploratory between-groups analysis will be performed at Day 31 using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates</li> <li>For Boostrix booster response to antigens PT, FHA and PRN, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately</li> </ul> |
| | Anti-D concentration Anti-T concentration | <ul> <li>The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for US and ex-US pooled data and separately</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-D, anti-Twill be calculated at Screening and Day 31 post vaccination for US and ex-US pooled data and separately.</li> <li>Protection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately.</li> </ul> |

209141 (RSV MAT-011)

Statistical Analysis Plan Amendment 4

# 9.1.1.1. Laboratory assays cut-offs for humoral immunity (Antibody determination) (Amended 03-DEC-2020)

A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay. The cut-off tests for immunogenicity evaluation will be as per following:

| Sample | Component | Method | Unit | Cut-off* | ULOQ |
|---|---|---|---|---|---|
| Serum | Respiratory Syncytial Virus A Ab neutralizing | NEU | ED60 and/or IU<br>(international unit) | 18 for ED60<br>56 for IU | ED60 : 123535<br>IU : 217400 |
| Serum | Respiratory Syncytial Virus<br>PreF3 Ab.lgG concentration | ELI | ELU/mL | 25 | 251 769 |
| Serum | Bordetella<br>pertussis.Filamentous<br>Hemaglutinin Ab.lgG | ELI | IU/mL | 2.046 | 3182.397 |
| Serum | Bordetella pertussis.Pertactin Ab.lgG | ELI | IU/mL | 2.187 | 6313.300 |
| Serum | Bordetella<br>pertussis.Pertussis Toxin<br>Ab.lgG | ELI | IU/mL | 2.693 | 883.559 |
| Serum | Corynebacterium<br>diphtheriae.Diphtheria Toxoid<br>Ab.lgG | ELI | IU/mL | 0.030 | 59.545 |
| Serum | Clostridium tetani.Tetanus<br>Toxoid Ab.lgG | ELI | IU/mL | 0.037 | 116.428 |

Ab = antibody; ELI = Enzyme-linked immunosorbent assay (ELISA); IgG = immunoglobulin G; RSV = respiratory syncytial virus; ED60 = serum dilution inducing 60% inhibition in plaque forming units; IU/ml = International units/milliliter, IU= International units

Assay cut-off and unit might be subject to change before starting of testing (e.g. in case of requalification, revalidation or standardisation). In this case, this will be documented in the clinical report.

# 9.2. Statistical Method

NA

# 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

# 10.1.2. Handling of missing data

## 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

# 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

## 10.1.2.3. Solicited adverse events (Amended 03-DEC-2020)

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited symptoms based on the Exposed
- Set Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after vaccination will be considered not having that symptom after vaccination.
  - When a specific solicited adverse event is marked as having not occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=N for the specified post-vaccination period for the adverse event in question), all daily measurements will be imputed as Grade 0.
  - When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.
  - When a specific solicited adverse event is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the adverse event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows, also counting this AE as "unknow" row of the solicited adverse event summary tables. Dose without symptom sheets documented will be excluded.

# 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

## 10.1.3. Data derivation

# 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

# 10.1.3.2. Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

# 10.1.3.3. Height

Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows:

Height in centimeters = Height in inches  $\times 2.54$ 

## 10.1.3.4. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (Weight in kilograms) / (Height in meters)<sup>2</sup>

# 10.1.3.5. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

# 10.1.3.6. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

# 10.1.3.7. Geometric mean titres (GMTs) and concentrations (GMCs)

Geometric Mean Titre (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Antibody titres or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

# 10.1.3.8. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

## 10.1.3.9. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited adverse event period.

# 10.1.3.10. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# 10.1.3.11. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a subject following multiple vaccines will be counted by as only one occurrence. However specific tables or figures could be conducted to report solicited local events by occurrence.

# 10.1.4. Display of decimals

# 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.
209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

## 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values are below 10kg where one decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with one decimal.

## 10.1.4.4. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| <b>GMT or GMC value</b> | Number of decimals to display |
|-------------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

#### 10.1.5. Statistical methodology

### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

209141 (RSV MAT-011) Statistical Analysis Plan Amendment 4

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Miettinen and Nurminen [Miettinen, 1985].

# 10.2. TFL TOC

The Table Figure Listing (TFL) Table of Content (TOC) which itemizes the planned list of TFL and their associated lay-out is developed as a separate document.

## 11. REFERENCES

Camargo ME, Silveira L, Furuta JA, Oliveira EP, Germek OA. Immunoenzymatic assay of anti-diphtheric toxin antibodies in human serum. *J Clin Microbiol*. 1984 Oct;20(4):772-4.

Christy C, Pichichero ME, Reed GF, Effect of Gender, Race, and Parental Education on Immunogenicity and Reported Reactogenicity of Acellular and Whole-Cell Pertussis Vaccines. Pediatrics (1995), 96(3)

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

Melville-Smith ME, Seagroatt VA, Watkins JT. A comparison of enzyme-linked immunosorbent assay (ELISA) with the toxin neutralization test in mice as a method for the estimation of tetanus antitoxin in human sera. *J Biol Stand*. 1983 Apr;11(2):137-44.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. Statistics in Medicine, 1985;4,213-226.

Vidor E, Plotkin SA. Immunogenicity of a two-component (PT & FHA) acellular pertussis vaccine in various combinations *Hum Vaccin*. 2008 Sep-Oct;4(5):328-40.

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | Phase II randomized, observer-blind, placebo-controlled, multi-country study in healthy non-pregnant women 18-45 years of age to evaluate the safety, reactogenicity and immunogenicity of a single intramuscular dose of GSK Biologicals' investigational RSV maternal vaccine (GSK388550A) when given alone and given in co-administration with a single intramuscular dose of Boostrix (US formulation SB776423 or ex-US formulation SB263855). |
| eTrack study number and<br>Abbreviated Title | 209141 (RSV MAT-011) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 21 October 2019 |
| <b>Date of Statistical Analysis</b> | Amendment 2 Final: 28 FEB 2020 |
| plan amendment | Amendment 3 Final: 03 April 2020 |
| APP 9000058193 | Statistical Analysis Plan Template V4 (Effective date: 3June2019) |

209141 (RSV MAT-011) Statistical Analysis Plan

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF A | ABBREVI | ATIONS | | 4 |
| 1. | DOC | JMENT H | ISTORY | | 7 |
| 2. | OBJE | CTIVES/ | ENDPOINTS | | 7 |
| 3. | STUE | DY DESIG | N | | 9 |
| 4. | ANAL | | | 3-APR-2020) | |
| | 4.1. | | | | |
| | | 4.1.1. | Exposed Set. | | 13 |
| | | 4.1.2. | | Analysis Set | |
| | 4.2. | Criteria | for eliminating o | data from Analysis Sets | 13 |
| | | 4.2.1. | | om Exposed Set (ES) | 13 |
| | | 4.2.2. | Elimination fro | om Per-protocol analysis Set (PPS) | 13 |
| | | | | cluded subjects from Per-protocol analysis | 14 |
| | | 4.2.3. | | om solicited safety set | |
| | | 7.2.0. | | cluded subjects | |
| | | | | 2.3.1.1. Solicited safety set | |
| 5. | STAT | | | | |
| | 5.1. | Demog | | | |
| | | 5.1.1. | Analysis of de | emographics/baseline characteristics planned | |
| | | | in the protoco | l <sup>*</sup> | 15 |
| | | 5.1.2. | Additional cor | nsiderations | 16 |
| | 5.2. | Immuno | genicity | | 17 |
| | | 5.2.1. | Analysis of im | munogenicity planned in the protocol | |
| | | | (Amended 03 | -APR-2020) | 17 |
| | | 5.2.2. | Additional cor | nsiderations | 18 |
| | | | | tween group analysis | |
| | | | | rcentage difference between two groups | |
| | 5.3. | Analysi | | eactogenicity | |
| | | 5.3.1. | | fety and reactogenicity planned in the | |
| | | | protocol (Ame | ended 03-APR-2020) | 20 |
| | | 5.3.2. | | nsiderations | |
| | | | | alysis of solicited events | |
| | | | | alysis of Unsolicited Adverse Events | |
| | | | | ombined Solicited and Unsolicited Adverse | |
| | | | | ents | 24 |
| | | | | her analysis | |
| 6. | ANAL | YSIS INT | ERPRETATION | <b>\</b> | 24 |
| _ | | | | | •- |
| 7. | | | | | |
| | 7.1. | | | | |
| | | 7.1.1. | | study | |
| | 7.2. | Statistic | al consideration | ns for interim analyses | 25 |

209141 (RSV MAT-011) Statistical Analysis Plan

| 8. | CHAN | IGES FRO | OM PLANNE | ED ANALYSES <i>(AMENDED 03-APR-2020)</i> | 26 |
|---|---|---|---|---|---|
| 9. | | | | ERIVATION RULES AND STATISTICAL | 26 |
| | 9.1. | | | | |
| | 9.1. | | | enicity (Amended 07-APR-2020) | |
| | | 9.1.1.1. | | / assays cut-offs for humoral immunity (Antibody | |
| | 9.2. | Ctatiation | | tion) (Amended 03-APR-2020) | |
| | 9.2. | Statistica | ai wethou | | 20 |
| 10. | ANNE | XES | | | 28 |
| | 10.1. | Business | s rules for st | tandard data derivations and statistical methods | 28 |
| | | 10.1.1. | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | 10.1.2.2. | Laboratory data | 29 |
| | | | | Solicited adverse events | |
| | | | | Unsolicited adverse events | |
| | | 10.1.3. | | ation | |
| | | | 10.1.3.1. | | |
| | | | 10.1.3.2. | | |
| | | | 10.1.3.3. | Height | |
| | | | 10.1.3.4. | | |
| | | | | Temperature | |
| | | | | Numerical serology results | |
| | | | 10.1.3.7. | | |
| | | | 10.1.0.7. | concentrations (GMCs) | 31 |
| | | | 10.1.3.8. | Onset day | 32 |
| | | | 10.1.3.0. | | |
| | | | | Counting rules for combining solicited and | 52 |
| | | | 10.1.5.10. | unsolicited adverse events | 33 |
| | | | 10 1 2 11 | Counting rules for occurrences of solicited | 32 |
| | | | 10.1.3.11. | adverse events | 22 |
| | | 10.1.4. | Display of | decimals | |
| | | 10.1.4. | | Percentages | |
| | | | | Differences in percentages | |
| | | | 10.1.4.2. | Corological summers statistics | 33 |
| | | 10 1 E | | Serological summary statistics | |
| | | 10.1.5. | | methodology | |
| | | | | Exact confidence intervals around proportions | 34 |
| | | | 10.1.5.2. | Standardized asymptotic confidence intervals | 0.4 |
| | 40.0 | TCL TO | _ | around differences in proportions | |
| | 10.2. | 1FL 100 | | | 34 |
| 11 | RFFF | RENCES | | | 35 |

209141 (RSV MAT-011) Statistical Analysis Plan

## LIST OF ABBREVIATIONS

**Ab** Antibody

**AE(s)** Adverse Event(s)

**AE** Adverse Event

Anti- Antibodies against

**BS H** Blood Sample Humoral

**CDC** Centers for Disease Control

CI Confidence Interval

CLS Clinical Laboratory Sciences

**CoP** Correlate of Protection

**D** Diphtheria

**dTpa** Diphtheria, Tetanus and acellular Pertussis

eCRF electronic Case Report Form

**ELISA** Enzyme-Linked Immunosorbent Assay

**EoS** End of Study

**eTDF** Electronic Temperature excursion Decision Form

**Ex-US** Outside the US

**FDA** Food and Drug Administration, United States of America

FHA Filamentous Hemagglutinin

FU Follow-up

**GCP** Good Clinical Practice

**GMC** Geometric Mean Concentration

**GMT** Geometric Mean Titer

**GSK** GlaxoSmithKline

**IAF** Informed Assent Form

209141 (RSV MAT-011) Statistical Analysis Plan

**IB** Investigator Brochure

ICF Informed Consent Form

**ICH:** International Council on Harmonisation

**IEC** Independent Ethics Committee

IgG Immunoglobulin

IM Intramuscular

IMP Investigational Medicinal Product

**IND** Investigational New Drug

**IRB** Institutional Review Board

**LAR** Legally Acceptable Representative

**LSLV** Last Subject Last Visit

MACDP Metropolitan Atlanta Congenital Defects Program

**MedDRA** Medical Dictionary for Regulatory Activities

**Nab** Neutralizing antibody

**PCD** Primary Completion Date

**PP** Per protocol

**PRN** Pertactin

**PRO** Patient Related Outcomes

PT Pertussis Toxoid

**RRA** Recruitment/Randomisation Agreement

**RSV** Respiratory Syncytial Virus

**RSVPreF3** RSV maternal vaccine

**SAE:** Serious Adverse Event

**SBIR** Source data Base for Internet Randomisation

**SD** Standard Deviation

209141 (RSV MAT-011) Statistical Analysis Plan

**SDV** Source Document Verification

**SmPC** Summary of Product Characteristics

**SPM** Study Procedures Manual

**SRT** Safety Review Team

T Tetanus

**UP** Urine Pregnancy Test

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|--------------------------|
| 03 APR 2020 | Amendment 3 | Amendment 3: 03-APR-2020 |
| 28 FEB 2020 | Amendment 2 | Amendment 2: 28-FEB-2020 |
| 21 Oct 2019 | first version | Final: 28 JUN 2019 |

# 2. OBJECTIVES/ENDPOINTS

Table 1 Study objectives and endpoints (Amended 03-APR-2020)

| Objectives | | | Endpoints |
|---|---|---|---|
| Primary (US + ex-U | | | a to be pooled) |
| Safe | ty | Safe | ty |
| • | To evaluate the safety and reactogenicity of 2 dose levels (60 and 120 $\mu g$ ) of RSVPreF3 when given alone or co-administered with dTpa from Vaccination up to Day 31. | | Occurrence of any Adverse Events (AEs) from Vaccination to Day 31: — Occurrence of each solicited local AEs at the site of injection in both limbs from Vaccination to Day 8; |
| | | | Occurrence of solicited general AEs from<br>Vaccination to Day 8; |
| | | | <ul> <li>Occurrence of any unsolicited AEs from<br/>Vaccination to Day 31;</li> </ul> |
| | | | <ul> <li>Occurrence of Serious Adverse Events (SAEs) from Vaccination to Day 31.</li> </ul> |
| Imm | unogenicity | Imm | unogenicity |
| • | To evaluate the humoral immune response to 2 dose levels (60 and 120 $\mu g)$ of RSVPreF3 when given alone and co-administered with dTpa, at Screening, Day 8 and Day 31. | • | RSV A neutralizing antibody titers at Screening,<br>Day 8 and Day 31 in all groups<br>RSV IgG antibody concentrations at Screening, Day<br>8 and Day 31. |
| | Secondary (US and ex-US data to be | e considered pooled, then separately) | |
| Safe | ty | Safe | ty |
| • | To evaluate the safety and reactogenicity of 2 dose levels (60 and 120 $\mu g$ ) of RSVPreF3 when given | | Occurrence of any AEs from Vaccination to Day 31, for all subjects: |
| | alone or co-administered with dTpa from Vaccination up to Day 31 by formulation. | | <ul> <li>Occurrence of each solicited local AE at the site<br/>of injection in both limbs from Vaccination to<br/>Day 8</li> </ul> |
| | | | <ul> <li>Occurrence of solicited general AEs from<br/>Vaccination to Day 8</li> </ul> |
| | | | <ul> <li>Occurrence of any unsolicited AEs from<br/>Vaccination to Day 31</li> </ul> |
| | | | <ul> <li>Occurrence of Serious Adverse Events (SAEs) from Vaccination to Day 31.</li> </ul> |
| • | To evaluate the safety of 2 dose levels (60 and 120 µg) of RSVPreF3 when given alone and co-administered with dTpa compared to dTpa-Placebo groups from Vaccination up to Day 181. | • | Occurrence of SAEs from Vaccination up to Day 181 |
| • | To evaluate the safety of 2 dose levels (60 and 120 $\mu$ g) of RSVPreF3 when given alone and coadministered from Vaccination up to Day 181. by formulation. | | Occurrence of SAEs from Vaccination up to Day 181 |

209141 (RSV MAT-011) Statistical Analysis Plan

| Occurrence of SAEs from Vaccination up to Day 181 nogenicity RSV A neutralizing antibody titers at Screening, Day |
|---|
| • , |
| RSV A neutralizing antihody titers at Screening, Day |
| 8, Day 31,. RSV IgG antibody concentrations at Screening, Day 8, Day 31. |
| Antibody concentrations against pertussis toxoid (anti-PT), filamentous hemagglutinin (anti-FHA), and pertactin (anti-PRN) concentrations at Screening and Day 31. |
| Anti-D concentrations at Screening and Day 31. |
| Anti-T concentrations at Screening and Day 31. |
| vaccination by formulation. Tertiary |

19-SEP-2019

be performed.

## 3. STUDY DESIGN

Figure 1 Study design overview (Amended 07-APR-2020)



Note: study groups labeled X = ex-US; study groups labeled U = US. V = visit, C = phone contact

= Vaccination; N = number of subjects; V = Visit; D = Day; AE = adverse event; UP = Urine pregnancy test; CHS = Chemical/Hematological Screening, FU = follow-up

BSH = blood sample (5 mL) for humoral immune responses (RSV-A neutralization and RSV IgG antibody concentrations at Screening, Visit 2 [Day 8] and Visit 3 [Day 31], and dTpa ELISAs at Screening and Visit 3 [Day 31])

The study will be conducted with 2 formulations of dTpa, dTpa\_300 (in the US) and dTpa\_500 (ex-US) [Christy, 1995].

Approximately 500 eligible subjects (250 in the US and 250 ex-US) will be enrolled. Of these, approximately 250 subjects will be randomized to 5 US study groups in a 1:1:1:1:1 ratio using SBIR, and the remaining approximately 250 will be randomized to 5 ex-US study groups in a 1:1:1:1:1 ratio using SBIR. The randomization algorithm will use a minimization procedure by treating study formulation (US and ex-US) as a stratification factor, and age at the time of vaccination (18-32 or 33-45 years of age) and center as minimization factors.

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements,

including those specified in the schedule of activities, are essential and required for study conduct.

- Type of study: self-contained
- **Experimental design:** multi-centric study, multi-country Phase II, observer-blind, randomized, with 5 parallel groups in each formulation (US, ex-US).
- **Duration of the study:** Approximately 6 months for each enrolled subject
  - Epoch 001: Screening
  - Epoch 002: Primary (i.e., vaccination phase) starting at Visit 1 (Day 1) and ending just before the Visit 3 (Day 31)
  - Epoch 003: Follow-up contact on Day 181
- Primary completion Date (PCD): Visit 3 (Day 31) or last visit of Primary Epoch
- End of Study (EoS): Last testing results released of samples collected at Visit 3, to occur no later than 8 months after last subject last visit (LSLV), which occurs with Contact 1 on Day 181.

## • Study groups:

Table2 Study groups, pooled study groups (Amended 03-APR-2020)

| Pooled Groups label in tables | Pooled definition for footnote | Group label in tables | Group definition for footnote |
|---|---|---|---|
| RSV120_dTpa | Subjects who received | XRSV120_dTpa | Subject who received RSV MAT 120 and<br>Boostrix-ex-US (dTpa_500) |
| 1101120_0100 | RSV120 and dTpa | URSV120_dTpa | Subjects who received RSV MAT 120 and<br>Boostrix-US (dTpa_300) |
| RSV120_Placebo | XPlacebo_R Subjects who received | | Subject who received RSV MAT 120 and Placebo |
| 1.67 120_1 145636 | RSV120 and placebo | UPlacebo_RSV120 | Subject who received RSV MAT 120 and Placebo |
| RSV60_ dTpa | Subjects who received | XRSV60_dTpa | Subjects who received RSV MAT 60 and<br>Boostrix-ex-US (dTpa_500) |
| | RSV60 and dTpa | URSV60_dTpa | Subjects who received RSV MAT 60 and<br>Boostrix-US (dTpa_300) |
| RSV60_Placebo | RSV60 Placebo Subjects who received | | Subjects who received RSV MAT 60 and Placebo |
| | RSV60 and placebo | UPlacebo_RSV60 | Subject who received RSV MAT 60 and Placebo |
| dTpa_Placebo | Subjects who received<br>Boostrix(dTpa) and | XPlacebo_dTpa | Subject who received <i>Boostrix</i> -ex-US (dTpa_500) and Placebo |
| , . <u></u> | Placebo | UPlacebo_dTpa | Subject who received <i>Boostrix</i> -US (dTpa_300) and Placebo |



Table 3 Study groups, treatment and epochs foreseen in the study (*Amended 03-APR-2020*)

| | Nemahan | A | | Epochs<br>(Blinding) | | |
|---|---|---|---|---|---|---|
| Study Groups | Number<br>of<br>subjects | Age<br>(Min-<br>Max) | Treatment<br>name | Epoch 001<br>(Screening) | Epoch 002<br>(observer-<br>blind) | Epoch<br>003<br>(single-<br>blind) |
| XRSV120_dTpa | 50 | 18 –<br>45<br>years | RSV MAT<br>120<br>Boostrix-ex-<br>US<br>(dTpa_500) | Х | x | х |
| Xplacebo_RSV120 | 50 | 18 –<br>45<br>years | RSV MAT<br>120<br>Placebo | Х | x | X |
| XRSV60_dTpa | 50 | 18 –<br>45<br>years | RSV MAT 60<br>Boostrix-ex-<br>US<br>(dTpa_500) | X | X | X |
| Xplacebo_RSV60 | 50 | 18 –<br>45<br>years | RSV MAT 60<br>Placebo | Х | x | X |
| Xplacebo_dTpa | 50 | 18 –<br>45<br>years | Boostrix-ex-<br>US<br>(dTpa_500)<br>Placebo | х | Х | Х |
| URSV120_dTpa | 50 | 18 –<br>45<br>years | RSV MAT<br>120<br>Boostrix-US<br>(dTpa_300) | X | Х | X |
| Uplacebo_RSV120 | 50 | 18 –<br>45<br>years | RSV MAT<br>120<br>Placebo | Х | Х | X |
| URSV60_dTpa | 50 | 18 –<br>45<br>years | RSV MAT 60<br>Boostrix-US | Х | Х | X |
| Uplacebo_RSV60 | 50 | 18 –<br>45<br>years | RSV MAT 60<br>Placebo | Х | Х | Х |
| Uplacebo_dTpa | 50 | 18 –<br>45<br>years | Boostrix-US<br>(dTpa_300)<br>Placebo | Х | Х | X |

209141 (RSV MAT-011) Statistical Analysis Plan

- Control: (active comparator).
- **Treatment allocation**: (randomised stratified).
- **Blinding:** As described in <u>Table 3</u>.
- **Data collection**: standardised Electronic Case Report Form (eCRF). Solicited symptoms will be collected using a subject paper Diary (pDiary).
- Safety monitoring:

If the investigator becomes aware of a holding rule being met, he/she will suspend vaccination and will inform GSK immediately.

## 4. ANALYSIS SETS (Amended 03-APR-2020)

### 4.1. Definition

For purposes of analysis, the following analysis sets are defined:

| Analysis Set | Description |
|---|---|
| Enrolled Subjects who agreed to participate in a clinical study after completion o informed consent process. And subject is not a screen failure. | |
| Exposed All subjects who received at least 1 dose of the study treatment. The allo in a group is done in function of the administered treatment. | |
| Per Protocol | All subjects who received at least 1 dose of the study treatment to which they are randomised and have post-vaccination data minus subjects with protocol deviations that lead to exclusion |
| Solicited Safety | All subjects who received at least 1 dose of the study treatment (Exposed Set) who have solicited safety data |

## 4.1.1. Exposed Set

The ES will include all subjects with study vaccine administration documented.

• A **safety** analysis based on the ES will include all vaccinated subjects.

## 4.1.2. Per Protocol Analysis Set

Per protocol analysis set will be defined by time points. It will include all of enrolled subjects who have immunogenicity data at Screening, Day 8 and Day 31.

• An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available, If, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

## 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES

## 4.2.2. Elimination from Per-protocol analysis Set (PPS)

Code 1030 (Study vaccine not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from PPS

## 4.2.2.1. Excluded subjects from Per-protocol analysis set

A subject will be excluded from the PPS analysis under the following conditions

Table 4 Elimination code and condition (*Amended 03-APR-2020*)

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 800 | Fraudulent data | All | All |
| 900 | Invalid informed consent | All | All |
| 1030 | Study vaccine not administered at all | All | Safety, immunogenicity |
| 1040.Vx+* | Administration of concomitant vaccine(s) forbidden in the protocol | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |
| 1050 | Randomisation failure | All | Immunogenicity |
| 1060 | Randomisation code was broken | All | Immunogenicity |
| 1070** | Subjects got vaccinated with the correct vaccine but containing an incorrect volume | All | Immunogenicity |
| 1070** | Vaccination not according to protocol (site of injection, route of administration, wrong replacement of study treatment administered) | All | Immunogenicity |
| 1070** | Study treatment not prepared as per protocol (e.g. reconstitution) | All | Immunogenicity |
| 1070** | Other deviations related to wrong study treatment/administration/dose | All | Immunogenicity |
| 1070** | Study treatment administered while contraindication | All | Immunogenicity |
| 1080 | Vaccine temperature deviation | All | Immunogenicity |
| 1090 | Expired vaccine administered | All | Immunogenicity |
| 2010 | Protocol violation (inclusion/exclusion criteria) DOB – VAC – 18-45 years | All | Immunogenicity |
| 2150 | Failure to report safety events per protocol | All | Safety |
| 2040.Vx+* | Administration of any medication forbidden by the protocol | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2040.Vx+* | Device, excluded by the protocol, was administered | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2050.Vx+* | Intercurrent medical conditions which are exclusionary as per protocol | Visit 3/Day 31 | Immunogenicity |
| 2060.Vx+* | Concomitant infection related to the vaccine which may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |
| 2070.Vx+* | Concomitant infection not related to the vaccine but may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181<br>Visit 4/Day 365 | Immunogenicity |

| Code | Condition under which the code is used | Visit (timepoints)<br>where the code is<br>applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 2090.Vx | Subjects did not comply with blood sample schedule: • For PPS at Day 8, check the interval from vaccination to day 8 BS = 7 – 10 days; • For PPS at Day 31, check the interval from vaccination to day 31 BS = 30 – 45 days; • For PPS at Day 181, check the interval from phone contact to visit 4 BS=0-30 days | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |
| 2100.Vx | Serological results not available post-vaccination | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |
| 2120.Vx | Obvious incoherence or abnormality or error in data | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |
| 2130.Vx | Testing performed on samples not aligned with ICF | Visit 2/Day 8<br>Visit 3/Day 31<br>Visit 4/Day 181 | Immunogenicity |

<sup>\*</sup>Attribution of these elimination codes to subject need CRDL review of individual listing

DOB-Date of Birth, VAC-Vaccination, BS- Blood Sample

## 4.2.3. Elimination from solicited safety set

## 4.2.3.1. Excluded subjects

## 4.2.3.1.1. Solicited safety set

Code 1030 (Study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used for identifying subjects eliminated from the solicited safety set.

## 5. STATISTICAL ANALYSES

## 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

These analyses will be performed on the Exposed set and on the Per protocol set for immunogenicity.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

Vx+ indicates subjects whose immunogenicity data will be eliminated from a specific visit onwards; Vx indicates subjects whose immunogenicity data will be eliminated from a specific visit.

209141 (RSV MAT-011) Statistical Analysis Plan

For all subjects, demographic characteristics (e.g., age at vaccination (18–32; 33-45 years), race and ethnicity, vaccination history will be summarized by overall and vaccine group using descriptive statistics.

- Frequency tables will be generated for categorical variables such as centre.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height, weight and body mass index (BMI).

## 5.1.2. Additional considerations

Demographic characteristics will also be summarized on Enrolled Set for web public disclosure.

Subject disposition will be summarized by group using descriptive statistics:

• Number of subjects screened, randomised, vaccinated and withdrawn including withdrawal reasons in each group and overall will be tabulated.

Vital signs will be summarized by group using descriptive statistics at all timepoint(s) the information is collected on Exposed Set and Per-protocol Set.

Summary of important protocol deviations leading to elimination will be tabulated by group. An individual listing will also be provided.

Summary of medical history will be performed on Exposed Set by Medical Dictionary for Regulatory Activities (MedDRA) and preferred term.

Summary of vaccination history will be performed on Exposed Set by using GSKDRUG dictionary.

Additional analyses by country and/or by site may be performed if deemed necessary

# 5.2. Immunogenicity

# 5.2.1. Analysis of immunogenicity planned in the protocol (*Amended 03-APR-2020*)

The primary analysis on immunogenicity will be based on the Per Protocol set. If, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more, a second analysis based on the Exposed Analysis Set will be performed to complement the Per Protocol analysis.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled) |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically pooled.</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI pooled.</li> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentrations may be calculated at</li> </ul> |
| | <ul> <li>Screening, and/or Day 8, and/or Day 31 pooled for all subjects.</li> <li>A further exploratory between-groups analysis will be performed at Day 8 or Day 31 using an ANCOVA model by including study groups, study formulation (US and ex-US), age category, and level of antibodies at Screening as covariates.</li> </ul> |

| Endpoint | Statistical Analysis Methods |
|---|---|
| Secondary | (US and ex-US data to be considered pooled, then separately |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | GMCs/GMTs and their 95% CI will be tabulated and represented graphically by formulation (US and ex-US). |
| | Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI by formulation (US and ex-US). |
| | Antibody titer/concentration will be displayed using reverse cumulative curves by formulation (US and ex-US). |
| | The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points by formulation (US and ex-US). |
| | <ul> <li>Response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by group for<br/>each formulation (US and ex-US).</li> </ul> |
| | Booster responses to PT, FHA and PRN antigens are defined as: |
| | <ol> <li>For subjects with pre-vaccination antibody concentration below the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the assay cut-offs,</li> </ol> |
| | <ol> <li>For subjects with pre-vaccination antibody concentration between the assay cut-offs and<br/>below 4 times the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the<br/>pre-vaccination antibody concentration, and</li> </ol> |
| | 3. For subjects with pre-vaccination antibody concentration ≥ 4 times the assay cut-offs: post-vaccination antibody concentration ≥ 2 times the pre-vaccination antibody concentration. |
| | <ul> <li>The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for each formulation (US and ex-US).</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-PT, anti-FHA, anti-PRN, anti-D, anti-T will be calculated at Screening and Day 31 pooled for all subjects and by formulation (US and ex-US).</li> </ul> |
| | <ul> <li>A further exploratory between-groups analysis in terms of anti-PT, anti-FHA, anti-PRN, anti-D, anti-T will be performed at Day 31 using an ANCOVA model by including study groups, study formulation (US and ex-US), age category, and level of antibodies at Screening as covariates.</li> </ul> |
| | • For Boostrix booster response to antigens PT, FHA and PRN, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group on Day 31 post vaccination will be calculated for each formulation. |
| | <ul> <li>For Boostrix seroprotection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for each formulation.</li> </ul> |
| Tertiary | Will be described in a Statistical Analysis Plan finalised before database unblinding/freezing. |

<sup>\*</sup>The statistical method will not be applied to primary endpoint. For detailed rationale, refer to Section 8.

\*\*pooled group definition is detailed in Table 2

#### 5.2.2. **Additional considerations**

At first analysis at Day 31 and final analysis at Day181, immunogenicity analysis will be performed on PPS.

## 5.2.2.1. Between group analysis

The Non-inferiority on RSV-A neutralizing antibody titers at 31 days post vaccination in the co-administration of RSVPre F3 vaccine + *Boostrix* compared to RSV+ Placebo will be evaluated based on the criterion below:

- The criterion to evaluate non-inferiority with respect to RSV-A neutralizing antibody titers is that the upper limits of the 95% CI on the GMT ratio (RSVPreF3 + *Placebo* divided by RSVPre3 + Boostrix) is less than or equal to 1.5 at 31 days post vaccination.

RSVPreF3 IgG antibody concentrations, RSV-A neutralizing antibody titers will applied to following model.

For the analysis of subjects at visit 3 (Day 31), the model will be explored and fitted via the procedure according to the following code:

```
PROC glm data=sero;
CLASS group;
MODEL log_val = baseline group age_cat country_US country_BE
Output out= pred;
LSMEANS group/pdiff cl alpha=0.1;
RUN:
```

where **log\_val** represents the log-transformed antibody value of the immunogenicity variable at a given post baseline timepoint (Day 8) or (Day 31), **baseline** is prevaccination logarithm10 transformation of the concentrations/titers, **group** indicates the study group, pooled groups (US and ex-US) will considered in model then separate by formulation. **age\_cat** is indicator variable (0/1) and will be treated as continuous in the model, age\_cat equals 0 if the age category at vaccination between 18 - 32 years, otherwise age\_cat equals 1 if age category is between 33 - 45 years at vaccination. **Country\_US** is indicator variable (0/1) and will treated as continuous in the model, if subject from US, then variable will equal to 1, otherwise equals to 0, **Country\_BE** is indicator variable (0/1) and will treated as continuous in model, if subject from BE, then variable equals to 1, otherwise equals to 0, if subject is from Canada, above two indicators equal to 0. The inclusion of age category at vaccination, in the model depends on the availability of the variable and the necessity, therefore, the above SAS code serves as a reference and may be adjusted according to the analysis needs.

When considering group as separated by Boostrix formulation, remove Country\_US and Country\_BE from model.\_

GMT/GMC ratios between vaccine groups obtained using above model will be calculated by exponentiating mean difference of logarithm- transformed titres. The 90% CI for GMT/GMC ratio will be obtained by exponential-transformation of the CI for the group least square mean of the log-transformed titres/concentration from the above model.

## 5.2.2.2. Percentage difference between two groups

We will conduct percentage difference of response rate in term of antigen PT, FHA and PRN [Camargo, 1984; Melville-Smith, 1983]. with the two-sided standardized asymptotic 95% CI in the RSVPreF3 dTpa group (minus) the dTpa Placebo group on Day 31.

Percentage difference of seroprotection rate in term of antigen D and antigen T [Vidor, 2008] with the two-sided standardized asymptotic 95% CI for RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group by formulation at Day 31 will be calculated.

# 5.3. Analysis of safety and reactogenicity

# 5.3.1. Analysis of safety and reactogenicity planned in the protocol (Amended 03-APR-2020)

The following safety analyses will be performed based on the Exposed Set. The following safety analysis will be performed on the pooled data then the US and ex-US separately.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled) |
| | The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any (solicited or unsolicited) AE during the 7-day or 30 day visit post vaccination period will be tabulated with exact 95% CI by study group. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits. |
| | The percentage of subjects reporting each individual solicited local AE (any related, any grade and grade 3 related AE and those resulting in medically attended visit) and solicited general AE (any related, any grade and grade 3 related AE and those resulting in medically attended visit) during the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) will be tabulated based on maximum intensity for each group. |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period will be tabulated for each group. Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | The percentage of subjects with any unsolicited AEs during the Day 1 to Day 30 follow-up period (i.e. on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term and SOC. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a CRDL and the signs |

209141 (RSV MAT-011) Statistical Analysis Plan

| Endpoint | Statistical Analysis Methods |
|---|---|
| | and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA SOC and Preferred Terms and reported during the 30-day follow-up period will be tabulated with exact 95% CI. SAEs will also be described in detail. |
| | The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period and during the 30-day follow-up period will be summarized by each group and pooled. |

209141 (RSV MAT-011) Statistical Analysis Plan

| Endpoint | Statistical Analysis Methods |
|---|---|
| Secondary | (US and ex-US data to be considered pooled, then separately) |
| | The percentage of subjects with at least one solicited AE(local and general), with at least one unsolicited AE and with any ("solicited or unsolicited") AE during the 7-day or 30 -day as well any SAE up to 180 days post vaccination will be tabulated with exact 95% CI by study group. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA SOC and Preferred Terms and reported during the 30-day follow-up period will be tabulated with exact 95% CI for each formulation (US and ex-US). |
| | The percentage of subjects reporting each individual solicited local AE (any grade, Grade 3 and those resulting in a medically attended visit) and solicited general AE (any grade, Grade 3, any related, Grade 3 related and those resulting in a medically attended visit) during the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) will be tabulated based on maximum intensity for each group for each formulation (US and ex-US). |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period will be tabulated for each group for each formulation (US and ex-US). Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | For each formulation (US and ex-US), the percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e. on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) SOC and preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| | The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) from vaccination up to day 30 will be summarized by each group for each formulation (US and ex-US). |
| Tertiary | Will be described in a Statistical Analysis Plan finalised before database unblinding/freezing. |

## 5.3.2. Additional considerations

# 5.3.2.1. Analysis of solicited events

The analysis of solicited events will be performed on Solicited Safety Set. The intensity of the following solicited events will be assessed as described:

Table 5 Intensity scales for solicited symptoms in adults

| Adults/Child (≥6 years) | | |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | CCI - This section collection questionn | ontained Clinical Outcome Assessment data aires or indices, which are protected by third and therefore have been excluded. |
| Redness at injection site | | |
| Swelling at injection site | | |
| Temperature* | | |
| Headache | | |
| Fatigue | | |
| Gastrointestinal symptoms<br>(nausea, vomiting, diarrhoea and/or<br>abdominal pain) | | |
| | | essment data collection questionnaires or t laws and therefore have been excluded. |

The maximum intensity of solicited administration site redness/swelling will be scored at GSK Biological as follows:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Duration in days of solicited local and general adverse events within 7 days after vaccination will be tabulated by study group and overall, and if needed by age group. The derivation rule of duration in days for solicited events is detailed in section 10.1.3.9.

## 5.3.2.2. Analysis of Unsolicited Adverse Events

The analysis of unsolicited events will be performed on Exposed Set.

#### 5.3.2.3. Combined Solicited and Unsolicited Adverse Events

The combined analysis of solicited and unsolicited events will be performed on Exposed Set. A summary of subjects with all combined solicited and unsolicited adverse events will be provided.

Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | Injection site pain | 10022086 |
| Redness | Redness at injection site | 10022098 |
| Swelling | Swelling at injection site | 10053425 |
| Fatigue | Fatigue | 10016256 |
| Fever | Fever | 10016558 |
| Headache | Headache | 10019211 |
| Gastrointestinal symptoms <sup>†</sup> | Gastrointestinal disorder | 10017944 |

Please note – to check for AE term in cDISC during dry run

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

## 5.3.2.4. Other analysis

Other safety analysis will be performed on Exposed Set.

Concomitant medications/products will be coded using the GSKDRUG dictionary. The number and percentage of subjects taking concomitant medications (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) within 7 days following vaccination, 30 days following vaccination and 12 months following vaccination will be summarized by group. A listing will also be provided.

## 6. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for most of these comparisons.

<sup>†</sup>Gastrointestinal symptoms include nausea, vomiting, diarrhoea and/or abdominal pain.

## 7. CONDUCT OF ANALYSES

## 7.1. Sequence of analyses

## 7.1.1. First and final study

Analyses to evaluate objectives and endpoints will be performed in steps.

A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints pertaining to safety and immunogenicity up to Day 31 are available. At this point, the statistician will be unblinded (i.e. individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblinded some specific subjects, the study will be considered as single-blind from this point onwards, with subjects and investigators remaining blinded up to study end. The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

The final end-of-study analysis will be performed when all data for at least primary and secondary endpoints up to study conclusion are available. Individual listings will only be provided at this stage. An integrated clinical study report containing all available data will be written and made available to the investigators.

The final study report will contain at least the final analyses of all primary and secondary endpoints. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These analyses will be documented in annex(es) to the study report and will be made available to the investigators at that time

| Description | Disclosure Purpose (CTRS=public posting, SR=study report, internal) |
|---|---|
| Final Analysis (E1_01) | Public disclosure, Study report |
| First Analysis (E1_02) | Public disclosure |

# 7.2. Statistical considerations for interim analyses

NA

# 8. CHANGES FROM PLANNED ANALYSES (AMENDED 03-APR-2020)

The calculation of GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3\_Placebo in terms of RSV-A Nab titers and RSV IgG antibody concentrations at Screening, Day 8 and Day 31 pooled for all subjects will be removedfrom analyses plan. We will report adjusted GMT/GMC ratio and their 95% CI which is generated from ANCOVA model

Adjusted GMT/GMC ratio with both 90% CI and 95% CI which are generated from ANCOVA model will be reported in terms of RSV-A Nab titers and RSV IgG antibody concentrations.

The calculation of GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa\_Placebo groups in terms of antigens PT, FHA, PRN, D and T will be added at Day 31 pooled for all RSV formulation.

Lab assay cut-off of RSV-A Nab titer for humoral immunity to be reported by using both IU/ml (International units/millilitre) and ED60

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section **** 

## 9.1. Data derivation

## 9.1.1. Immunogenicity (Amended 07-APR-2020)

For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

- For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude subjects with a missing or non-evaluable measurement.
- For the between group assessments, statistical model will be fitted based on the subjects having a result at both the baseline and the considered timepoint.

Following table will demonstrate all antigens will be analysed at considered time point for different treatment groups

| Immunogenicity<br>Endpoints | | Statistical Analysis Methods |
|---|---|---|
| RSVPreF3 IgG antibody concentration, and Neutralizing antibody titers against RSV-A RSVPreF3 | | <ul> <li>(US and ex-US data to be considered pooled, then separately)</li> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI</li> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> <li>A further exploratory between-groups of RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentration, analysis will be performed at Day 8 and Day 31 using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates</li> </ul> |
| Boostrix<br>(dTpa) | Booster response to PT Booster response to FHA Booster response to PRN | <ul> <li>For the subjects received RSVPreF3 dTpa and subjects received dTpa placebo</li> <li>Booster response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by group for US and ex-US pooled formulation and separately.</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-PT, anti-FHA, anti-PRN will be calculated between Day 31 over Screening for US and ex-US pooled data and separately.</li> <li>A further exploratory between-groups analysis will be performed at Day 31 using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates</li> <li>For Boostrix booster response to antigens PT, FHA and PRN, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately</li> </ul> |
| | Anti-D concentration Anti-T concentration | For the subjects received RSVPreF3 dTpa and subjects received dTpa placebo • The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for US and ex-US pooled data and separately • The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-D, anti-Twill be calculated at Screening and Day 31 for US and ex-US pooled data and separately. • Protection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately. |

# 9.1.1.1. Laboratory assays cut-offs for humoral immunity (Antibody determination) (Amended 03-APR-2020)

A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay. The cut-off tests for immunogenicity evaluation will be as per following:

| Sample | Component | Method | Unit | Cut-off* | ULOQ |
|---|---|---|---|---|---|
| Serum | Respiratory Syncytial Virus A<br>Ab neutralizing | NEU | ED60 and/or IU<br>(international unit) | 18 for ED60<br>56 for IU | ED60 : 123535<br>IU : 217400 |
| Serum | Respiratory Syncytial Virus<br>PreF3 Ab.lgG concentration | ELI | ELU/mL | 25 | 251 769 |
| Serum | Bordetella<br>pertussis.Filamentous<br>Hemaglutinin Ab.lgG | ELI | IU/mL | 2.046 | 3182.397 |
| Serum | Bordetella pertussis.Pertactin<br>Ab.lgG | ELI | IU/mL | 2.187 | 6313.300 |
| Serum | Bordetella<br>pertussis.Pertussis Toxin<br>Ab.lgG | ELI | IU/mL | 2.693 | 883.559 |
| Serum | Corynebacterium<br>diphtheriae.Diphtheria Toxoid<br>Ab.lgG | ELI | IU/mL | 0.030 | 59.545 |
| Serum | Clostridium tetani.Tetanus<br>Toxoid Ab.lgG | ELI | IU/mL | 0.037 | 116.428 |

Ab = antibody; ELI = Enzyme-linked immunosorbent assay (ELISA); IgG = immunoglobulin G; RSV = respiratory syncytial virus; ED60 = serum dilution inducing 60% inhibition in plaque forming units; IU/ml = International units/milliliter, IU= International units

Assay cut-off and unit might be subject to change before starting of testing (e.g. in case of requalification, revalidation or standardisation). In this case, this will be documented in the clinical report.

### 9.2. Statistical Method

NA

### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section **** (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Solicited adverse events

- For a given subject and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited symptoms based on the Exposed Set Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after vaccination will be considered not having that symptom after vaccination.
  - When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.
  - When a specific solicited adverse event is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified postvaccination period for the adverse event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited adverse event summary tables.
  - Dose without symptom sheets documented will be excluded.

#### 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

### 10.1.3. Data derivation

## 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

#### 10.1.3.2. Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

### 10.1.3.3. Height

Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows:

Height in centimeters = Height in inches  $\times 2.54$ 

### 10.1.3.4. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (Weight in kilograms) / (Height in meters) $^2$ 

## 10.1.3.5. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

## 10.1.3.6. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

## 10.1.3.7. Geometric mean titres (GMTs) and concentrations (GMCs)

Geometric Mean Titre (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Antibody titres or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

### 10.1.3.8. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.9. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited adverse event period.

## 10.1.3.10. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

## 10.1.3.11. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a subject following multiple vaccines will be counted by as only one occurrence. However specific tables or figures could be conducted to report solicited local events by occurrence

## 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

209141 (RSV MAT-011) Statistical Analysis Plan

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values are below 10kg where one decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with one decimal.
#### 10.1.4.4. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

# 10.1.5. Statistical methodology

#### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [, 1934].

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Miettinen and Nurminen [, 1985].

#### 10.2. TFL TOC

The Table Figure Listing (TFL) Table of Content (TOC) which itemizes the planned list of TFL and their associated lay-out is developed as a separate document.

## 11. REFERENCES

Camargo ME, Silveira L, Furuta JA, Oliveira EP, Germek OA. Immunoenzymatic assay of anti-diphtheric toxin antibodies in human serum. *J Clin Microbiol*. 1984 Oct;20(4):772-4.

Christy C, Pichichero ME, Reed GF, Effect of Gender, Race, and Parental Education on Immunogenicity and Reported Reactogenicity of Acellular and Whole-Cell Pertussis Vaccines. Pediatrics (1995), 96(3)

Melville-Smith ME, Seagroatt VA, Watkins JT. A comparison of enzyme-linked immunosorbent assay (ELISA) with the toxin neutralization test in mice as a method for the estimation of tetanus antitoxin in human sera. *J Biol Stand*. 1983 Apr;11(2):137-44.

Vidor E, Plotkin SA. Immunogenicity of a two-component (PT & FHA) acellular pertussis vaccine in various combinations *Hum Vaccin*. 2008 Sep-Oct;4(5):328-40.

# Signature Page for $\,209141$ TMF-1765379 $\,v1.0$

| Reason for signing: Approved | Name: Feng Gao |
|---|---|
| | Role: Approver |
| | Date of signature: 30-Apr-2020 16:03:07 GMT+0000 |

Signature Page for TMF-1765379 v1.0

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | Phase II randomized, observer-blind, placebo-controlled, multi-country study in healthy non-pregnant women 18-45 years of age to evaluate the safety, reactogenicity and immunogenicity of a single intramuscular dose of GSK Biologicals' investigational RSV maternal vaccine (GSK388550A) when given alone and given in co-administration with a single intramuscular dose of Boostrix (US formulation SB776423 or ex-US formulation SB263855). |
| eTrack study number and<br>Abbreviated Title | 209141 (RSV MAT-011) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 21 October 2019 |

APP 9000058193 Statistical Analysis Plan Template V4 (Effective date: 3June2019)

209141 (RSV MAT-011) Statistical Analysis Plan

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF A | ABBREVI | ATIONS | | 6 |
| 1. | DOC | JMENT H | IISTORY | | 9 |
| 2. | OBJE | CTIVES/ | ENDPOINTS | <b>.</b> | 9 |
| 3. | STUE | Y DESIG | :N | | 11 |
| 4. | | | | | |
| | 4.1. | | | | |
| | | 4.1.1. | | Set | |
| | | 4.1.2. | | col Analysis Set | |
| | 4.2. | | for eliminatin | ng data from Analysis Sets | 14 |
| | | 4.2.1. | Elimination | n from Exposed Set (ES) | 14 |
| | | 4.2.2. | Eliminatior 4.2.2.1. | from Per-protocol analysis Set (PPS)<br>Excluded subjects from Per-protocol analysis | |
| | | 4.0.0 | <b>-</b> 0 | set | |
| | | 4.2.3. | | from solicited safety set | |
| | | | 4.2.3.1. | Excluded subjects | |
| | | | | 4.2.3.1.1. Solicited safety set | 16 |
| 5. | STAT | | | | |
| | 5.1. | Demog | raphy | | 17 |
| | | 5.1.1. | Analysis of in the proto | f demographics/baseline characteristics planned | 17 |
| | | 5.1.2. | | considerations | |
| | 5.2. | _ | | | |
| | O. <b>_</b> . | 5.2.1. | | f immunogenicity planned in the protocol | |
| | | 5.2.2. | | considerations | |
| | | 0.2.2. | 5.2.2.1. | Between group analysis | |
| | | | 5.2.2.2. | Percentage difference between two groups | |
| | 5.3. | Analysi | | nd reactogenicity | |
| | 0.0. | 5.3.1. | Analysis o | f safety and reactogenicity planned in the | |
| | | 5.3.2. | Additional | considerations | 20 |
| | | J.J.Z. | 5.3.2.1. | | |
| | | | | Analysis of solicited events | |
| | | | 5.3.2.2.<br>5.3.2.3. | Analysis of Unsolicited Adverse Events Combined Solicited and Unsolicited Adverse | 23 |
| | | | | Events | <mark>23</mark> |
| | | | 5.3.2.4. | Other analysis | |
| 6. | ANAL | YSIS INT | ERPRETAT | ION | 24 |
| 7. | CONI | OUCT OF | ANAI YSES | | 24 |
| ٠. | 7.1. | | | es | |
| | 7.1. | 7.1.1. | | inal study | |
| | 72 | | | tions for interim analyses | 24 |

209141 (RSV MAT-011) Statistical Analysis Plan

| 8. | CHAN | IGES FRO | OM PLANNE | ED ANALYSES | 25 |
|---|---|---|---|---|---|
| 9. | | | | ERIVATION RULES AND STATISTICAL | 25 |
| | w∟17<br>9.1. | | | | |
| | 9.1. | | | | |
| | | 9.1.1.<br>9.1.1.1. | Laboratory | enicity<br>y assays cut-offs for humoral immunity (Antibody | |
| | 0.0 | Ctatiatia | | tion) | |
| | 9.2. | Statistica | ai ivietnod | | 27 |
| 10 | ANNE | XFS | | | 27 |
| | 10.1. | | | tandard data derivations and statistical methods | |
| | | | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | 0 | Laboratory data | |
| | | | 10.1.2.3. | Unsolicited adverse events | |
| | | 10.1.3. | | ation | |
| | | 10.1.0. | 10.1.3.1. | | |
| | | | | Weight | |
| | | | 10.1.3.2. | Height | |
| | | | 10.1.3.3. | Body mass index (BMI) | |
| | | | 10.1.3.4. | | |
| | | | 10.1.3.5. | Temperature | |
| | | | | Numerical serology results | 30 |
| | | | 10.1.3.7. | Geometric mean titres (GMTs) and | 20 |
| | | | 40 4 0 0 | concentrations (GMCs) | |
| | | | 10.1.3.8. | Onset day | |
| | | | 10.1.3.9. | | 30 |
| | | | 10.1.3.10. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 30 |
| | | | 10.1.3.11. | Counting rules for occurrences of solicited | |
| | | | | adverse events | |
| | | 10.1.4. | | decimals | |
| | | | 10.1.4.1. | | |
| | | | 10.1.4.2. | Differences in percentages | 32 |
| | | | 10.1.4.4. | Serological summary statistics | 32 |
| | | 10.1.5. | Statistical | methodology | |
| | | | | Exact confidence intervals around proportions | |
| | | | | Standardized asymptotic confidence intervals | |
| | | | | around differences in proportions | 33 |
| | 10.2. | TFL TO | J | around directorices in propertions | |
| | 3 | | | | |
| 11 | RFFF | RENCES. | | | 34 |

209141 (RSV MAT-011) Statistical Analysis Plan

# **LIST OF TABLES**

| | | PAGE |
|---------|----------------------------------------------------------|------|
| Table 1 | Study objectives and endpoints | 9 |
| Table 2 | Study groups, pooled study groups | 12 |
| Table 3 | Study groups, treatment and epochs foreseen in the study | 13 |
| Table 4 | Elimination code and condition | 15 |
| Table 5 | Intensity scales for solicited symptoms in adults | 22 |

209141 (RSV MAT-011) Statistical Analysis Plan

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 11 |

209141 (RSV MAT-011) Statistical Analysis Plan

# LIST OF ABBREVIATIONS

**Ab** Antibody

**AE(s)** Adverse Event(s)

**AE** Adverse Event

Anti- Antibodies against

**BS H** Blood Sample Humoral

**CDC** Centers for Disease Control

CI Confidence Interval

CLS Clinical Laboratory Sciences

**CoP** Correlate of Protection

**D** Diphtheria

dTpa Diphtheria, Tetanus and acellular Pertussis

eCRF electronic Case Report Form

**ELISA** Enzyme-Linked Immunosorbent Assay

**EoS** End of Study

eTDF Electronic Temperature excursion Decision Form

**Ex-US** Outside the US

**FDA** Food and Drug Administration, United States of America

**FHA** Filamentous Hemagglutinin

FU Follow-up

**GCP** Good Clinical Practice

**GMC** Geometric Mean Concentration

**GMT** Geometric Mean Titer

**GSK** GlaxoSmithKline

**IAF** Informed Assent Form

209141 (RSV MAT-011) Statistical Analysis Plan

**IB** Investigator Brochure

**ICF** Informed Consent Form

**ICH:** International Council on Harmonisation

**IEC** Independent Ethics Committee

IgG Immunoglobulin

IM Intramuscular

IMP Investigational Medicinal Product

**IND** Investigational New Drug

**IRB** Institutional Review Board

LAR Legally Acceptable Representative

LSLV Last Subject Last Visit

MACDP Metropolitan Atlanta Congenital Defects Program

**MedDRA** Medical Dictionary for Regulatory Activities

Nab Neutralizing antibody

**PCD** Primary Completion Date

**PP** Per protocol

**PRN** Pertactin

**PRO** Patient Related Outcomes

PT Pertussis Toxoid

**RRA** Recruitment/Randomisation Agreement

**RSV** Respiratory Syncytial Virus

**RSVPreF3** RSV maternal vaccine

**SAE:** Serious Adverse Event

**SBIR** Source data Base for Internet Randomisation

**SD** Standard Deviation

209141 (RSV MAT-011) Statistical Analysis Plan

**SDV** Source Document Verification

**SmPC** Summary of Product Characteristics

**SPM** Study Procedures Manual

**SRT** Safety Review Team

T Tetanus

**UP** Urine Pregnancy Test

# 1. DOCUMENT HISTORY

| Date Description | | Protocol Version |
|------------------|---------------|--------------------|
| 21 Oct 2019 | first version | Final: 28 JUN 2019 |

# 2. OBJECTIVES/ENDPOINTS

# Table 1 Study objectives and endpoints

| Objectives | Endpoints |
|---|---|
| Primary (US + ex-U | JS data to be pooled) |
| Safety | Safety |
| • To evaluate the safety and reactogenicity of 2 dose levels (60 and 120 μg) of RSVPreF3 when given alone or co-administered with dTpa from Vaccination up to Day 31. | Occurrence of any Adverse Events (AEs) from Vaccination to Day 31: Occurrence of each solicited local AEs at the site of injection in both limbs from Vaccination to Day 8; Occurrence of solicited general AEs from Vaccination to Day 8; Occurrence of any unsolicited AEs from Vaccination to Day 31; Occurrence of Serious Adverse Events (SAEs) from Vaccination to Day 31. |
| Immunogenicity | Immunogenicity |
| To evaluate the humoral immune response to 2 dose levels (60 and 120 μg) of RSVPreF3 when given alone and co-administered with dTpa, at Screening, Day 8 and Day 31. | <ul> <li>RSV A neutralizing antibody titers at Screening,<br/>Day 8 and Day 31 in all groups</li> <li>RSV IgG antibody concentrations at Screening, Day 8 and Day 31.</li> </ul> |
| Secondary (US and ex-US data to b | pe considered pooled, then separately) |
| Safety | Safety |
| <ul> <li>To evaluate the safety and reactogenicity of 2 dose<br/>levels (60 and 120 μg) of RSVPreF3 when given<br/>alone or co-administered with dTpa from Vaccination<br/>up to Day 31 by formulation.</li> </ul> | Occurrence of any AEs from Vaccination to Day 31, for all subjects: Occurrence of each solicited local AE at the site of injection in both limbs from Vaccination to Day 8 Occurrence of solicited general AEs from Vaccination to Day 8 Occurrence of any unsolicited AEs from Vaccination to Day 31 Occurrence of Serious Adverse Events (SAEs) from Vaccination to Day 31. |
| <ul> <li>To evaluate the safety of 2 dose levels (60 and<br/>120 μg) of RSVPreF3 when given alone and co-<br/>administered with dTpa compared to dTpa-Placebo<br/>groups from Vaccination up to Day 181.</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |
| <ul> <li>To evaluate the safety of 2 dose levels (60 and<br/>120 μg) of RSVPreF3 when given alone and co-<br/>administered from Vaccination up to Day 181 by<br/>formulation.</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |
| <ul> <li>To evaluate the safety of RSVPreF3 (pooled for all<br/>groups receiving RSVPreF3).</li> </ul> | Occurrence of SAEs from Vaccination up to Day<br>181. |

209141 (RSV MAT-011) Statistical Analysis Plan

| Objectives | Endpoints |
|---|---|
| Immunogenicity | Immunogenicity |
| <ul> <li>To evaluate the humoral immune response to 2<br/>dose levels (60 and 120 μg) of RSVPreF3 when<br/>given alone and co-administered with dTpa at<br/>Screening, Day 8 and Day 31 post vaccination by<br/>formulation.</li> </ul> | <ul> <li>RSV A neutralizing antibody titers at Screening, Day 8 and Day 31.</li> <li>RSV IgG antibody concentrations at Screening, Day 8 and Day 31.</li> </ul> |
| <ul> <li>To evaluate the humoral immune response to the<br/>pertussis component of the dTpa vaccine when<br/>given alone and co-administered with 2 dose levels<br/>(60 and 120 µg) of RSVPreF3 at Screening and Day<br/>31 by formulation.</li> </ul> | <ul> <li>Antibody concentrations against pertussis toxoid<br/>(anti-PT), filamentous hemagglutinin (anti-FHA), and<br/>pertactin (anti-PRN) concentrations at Screening<br/>and Day 31.</li> </ul> |
| <ul> <li>To evaluate the humoral immune response to the<br/>diphtheria (D) component of dTpa vaccine when<br/>given alone and co-administered with 2 dose levels<br/>(60 and 120 µg) of RSVPreF3 at Screening and Day<br/>31 post vaccination by formulation.</li> </ul> | Anti-D concentrations at Screening and Day 31. y |
| • To evaluate the humoral immune response to the tetanus (T) component of dTpa vaccine when given alone and co-administered with 2 dose levels (60 and 120 µg) of RSVPreF3 at Screening and Day 31 post vaccination by formulation. | |
| Tertiary | |
| If necessary, additional testing to further characterize the response to the RSV maternal investigational vaccine will be performed. | |

#### STUDY DESIGN

Figure 1 Study design overview



Note: study groups labeled X = ex-US; study groups labeled U = US.

= Vaccination; N = number of subjects; CHS= Chemical/Hematological Screening Visit; D = Day; AE = adverse event; UP = Urine pregnancy test; FU = follow-up; BSH = blood sample (5 mL) for humoral immune responses (RSV-A neutralization and RSV IgG antibody concentrations at Screening, Visit 2 [Day 8] and Visit 3 [Day 31], and dTpa ELISAs at Screening and Visit 3 [Day 31])

The study will be conducted with 2 formulations of dTpa, dTpa\_300 (in the US) and dTpa\_500 (ex-US) [Christy, 1995].

Approximately 500 eligible subjects (250 in the US and 250 ex-US) will be enrolled. Of these, approximately 250 subjects will be randomized to 5 US study groups in a 1:1:1:1:1 ratio using SBIR, and the remaining approximately 250 will be randomized to 5 ex-US study groups in a 1:1:1:1:1 ratio using SBIR. The randomization algorithm will use a minimization procedure by treating study formulation (US and ex-US) as a stratification factor, and age at the time of vaccination (18-32 or 33-45 years of age) and center as minimization factors.

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the schedule of activities, are essential and required for study conduct.

- Type of study: self-contained
- **Experimental design:** multi-centric study, multi-country Phase II, observer-blind, randomized, with 5 parallel groups in each formulation (US, ex-US).
- **Duration of the study:** Approximately 6 months for each enrolled subject
  - Epoch 001: Screening
  - Epoch 002: Primary (i.e., vaccination phase) starting at Visit 1 (Day 1) and ending just before the Visit 3 (Day 31)
  - Epoch 003: Follow-up contact on Day 181
- Primary completion Date (PCD): Visit 3 (Day 31) or last visit of Primary Epoch
- End of Study (EoS): Last testing results released of samples collected at Visit 3, to occur no later than 8 months after last subject last visit (LSLV), which occurs with Contact 1 on Day 181.
- Study groups:

Table 2 Study groups, pooled study groups

| Group<br>order | Group label | Group definition | Pooled Group<br>label | Pooled group definition |
|---|---|---|---|---|
| 1 | XRSV120_dTpa | Subject who received RSV<br>MAT 120<br>Boostrix-ex-US (dTpa_500) | RSV120_dTpa | Subjects who received RSV120 and dTpa |
| 2 | URSV120_dTpa | Subjects who received RSV<br>MAT 120<br>Boostrix-US (dTpa_300) | RSV120_dTpa | Subjects who received RSV120 and dTpa |
| 3 | XPlacebo_RSV120 | Subject who received RSV<br>MAT 120<br>Placebo | RSV120_Placebo | Subjects who received RSV120 and placebo |
| 4 | UPlacebo_RSV120 | Subject who received <i>RSV MAT 120</i> Placebo | RSV120_Placebo | Subjects who received RSV120 and placebo |
| 5 | XRSV60_<br>dTpa | Subjects who received RSV<br>MAT 60<br>Boostrix-ex-US (dTpa_500) | RSV60_dTpa | Subjects who received RSV60 and dTpa |
| 6 | URSV60_<br>dTpa | RSV MAT 60<br>Boostrix-US (dTpa_300) | RSV60_dTpa | Subjects who received RSV60 and dTpa |
| 7 | XPlacebo_RSV60 | Subjects who received RSV<br>MAT 60<br>Placebo | RSV60_Placebo | Subjects who received RSV60 and placebo |
| 8 | UPlacebo_RSV60 | Subject who received RSV MAT 60 Placebo | RSV60_Placebo | Subjects who received RSV60 and placebo |
| 9 | XPlacebo_dTpa | Subject who received<br>Boostrix-US (dTpa_500)<br>Placebo | dTpa_Placebo | Subjects who received Boostrix(dTpa) and Placebo |

209141 (RSV MAT-011) Statistical Analysis Plan

| Group order | Group label | Group definition | Pooled Group label | Pooled group definition |
|---|---|---|---|---|
| 10 | UPlacebo_dTpa | Subject who received Boostrix-US (dTpa_300) Placebo | dTpa_Placebo | Subjects who received Boostrix(dTpa) and Placebo |

Table 3 Study groups, treatment and epochs foreseen in the study

| | Nombonet | Age | | Epochs<br>(Blinding) | | |
|---|---|---|---|---|---|---|
| Study Groups | Number of subjects | (Min-<br>Max) | Treatment name | Epoch 001<br>(Screening) | Epoch 002<br>(observer-<br>blind) | Epoch 003<br>(single-<br>blind) |
| XRSV120_dTpa | 50 | 18 - 45<br>years | RSV MAT 120<br>Boostrix-ex-US<br>(dTpa_500) | Х | х | х |
| XPlacebo_RSV120 | 50 | 18 - 45<br>years | RSV MAT 120<br>Placebo | Х | х | х |
| XRSV60_dTpa | 50 | 18 - 45<br>years | RSV MAT 60<br>Boostrix-ex-US<br>(dTpa_500) | х | х | х |
| XPlacebo_RSV60 | 50 | 18 - 45<br>years | RSV MAT 60<br>Placebo | х | х | х |
| XPlacebo_dTpa | 50 | 18 - 45<br>years | Boostrix-ex-US<br>(dTpa_500)<br>Placebo | х | х | х |
| URSV120_dTpa | 50 | 18 – 45<br>years | RSV MAT 120<br>Boostrix-US<br>(dTpa_300) | Х | х | х |
| UPlacebo_RSV120 | 50 | 18 – 45<br>years | RSV MAT 120<br>Placebo | х | х | х |
| URSV60_dTpa | 50 | 18 - 45<br>years | RSV MAT 60<br>Boostrix-US | х | х | х |
| UPlacebo_RSV60 | 50 | 18 - 45<br>years | RSV MAT 60<br>Placebo | х | х | х |
| UPlacebo_dTpa | 50 | 18 – 45<br>years | Boostrix-US<br>(dTpa_300)<br>Placebo | Х | х | х |

- Control: (active comparator).
- Treatment allocation: (randomised stratified).
- **Blinding:** As described in Table 3
- **Data collection**: standardised Electronic Case Report Form (eCRF). Solicited symptoms will be collected using a subject paper Diary (pDiary).
- Safety monitoring:

If the investigator becomes aware of a holding rule being met, he/she will suspend vaccination and will inform GSK immediately.

#### 4. ANALYSIS SETS

#### 4.1. Definition

For purposes of analysis, the following analysis sets are defined:

| Analysis Set | Description |
|---|---|
| Enrolled | All subjects who completed the informed consent process and signed the informed consent form |
| Exposed | All subjects who received at least 1 dose of the study treatment. The allocation in a group is done in function of the administered treatment. |
| Per Protocol | All subjects who received at least 1 dose of the study treatment to which they are randomised and have post-vaccination data minus subjects with protocol deviations that lead to exclusion |
| Solicited Safety | All subjects who received at least 1 dose of the study treatment (Exposed Set) who have solicited safety data |

# 4.1.1. Exposed Set

The ES will include all subjects with study vaccine administration documented.

• A **safety** analysis based on the ES will include all vaccinated subjects.

# 4.1.2. Per Protocol Analysis Set

Per protocol analysis set will be defined by time points. It will include all of enrolled subjects who have immunogenicity data at Screening, Day 8 and Day 31.

• An **immunogenicity** analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available, If, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

## 4.2.2.1. Excluded subjects from Per-protocol analysis set

A subject will be excluded from the PPS analysis under the following conditions

Table 4 Elimination code and condition

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the code is<br>applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 800 | Fraudulent data | All | All |
| 900 | Invalid informed consent | All | All |
| 1030 | Study vaccine not administered at all | All | Safety, immunogenicity |
| 1040.Vx+* | Administration of concomitant vaccine(s) forbidden in the protocol | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 1050 | Randomisation failure | All | Immunogenicity |
| 1060 | Randomisation code was broken | All | Immunogenicity |
| 1070** | Subjects got vaccinated with the correct vaccine but containing an incorrect volume | All | Immunogenicity |
| 1070** | Vaccination not according to protocol (site of injection, route of administration, wrong replacement of study treatment administered) | All | Immunogenicity |
| 1070** | Study treatment not prepared as per protocol (e.g. reconstitution) | All | Immunogenicity |
| 1070** | Other deviations related to wrong study treatment/administration/dose | All | Immunogenicity |
| 1070** | Study treatment administered while contraindication | All | Immunogenicity |
| 1080 | Vaccine temperature deviation | All | Immunogenicity |
| 1090 | Expired vaccine administered | All | Immunogenicity |
| 2010 | Protocol violation<br>(inclusion/exclusion criteria)<br>DOB – VAC – 18-45 years | All | Immunogenicity |
| 2040.Vx+* | Administration of any medication forbidden by the protocol | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2040.Vx+* | Device, excluded by the protocol, was administered | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |

209141 (RSV MAT-011) Statistical Analysis Plan

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the code is<br>applicable | Applicable for analysis set/endpoint |
|---|---|---|---|
| 2050.Vx+* | Intercurrent medical conditions which are exclusionary as per protocol | Visit 3/Day 31 | Immunogenicity |
| 2060.Vx+* | Concomitant infection related to the vaccine which may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2070.Vx+* | Concomitant infection not related to the vaccine but may influence immune response | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2090.Vx | Subjects did not comply with blood sample schedule: • For PPS at Day 8, check the interval from vaccination to day 8 BS = 7 - 10 days; • For PPS at Day 31, check the interval from vaccination to day 31 BS = 30 - 45 days; | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2100.Vx | Serological results not available post-vaccination | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2120.Vx | Obvious incoherence or abnormality or error in data | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |
| 2130.Vx | Testing performed on samples not aligned with ICF | Visit 2/Day 8<br>Visit 3/Day 31 | Immunogenicity |

<sup>\*</sup>Attribution of these elimination codes to subject need CRDL review of individual listing

DOB-Date of Birth, VAC-Vaccination, BS- Blood Sample

# 4.2.3. Elimination from solicited safety set

## 4.2.3.1. Excluded subjects

#### 4.2.3.1.1. Solicited safety set

Code 1030 (Study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used for identifying subjects eliminated from the solicited safety set.

<sup>\*\*</sup> Attribution of code 1070 to a subject requires CRDL confirmation

Vx+ indicates subjects whose immunogenicity data will be eliminated from a specific visit onwards; Vx indicates subjects whose immunogenicity data will be eliminated from a specific visit.

#### 5. STATISTICAL ANALYSES

That standard data derivation rules and stat methods are described in section 10 while the study specific data derivation rules and stat methods are described in section 9

# 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

These analyses will be performed on the Exposed set and on the Per protocol set for immunogenicity.

For all subjects, demographic characteristics (e.g., age at vaccination (18 - 32; 33-45) years), race and ethnicity, vaccination history will be summarized by overall and vaccine group using descriptive statistics.

- Frequency tables will be generated for categorical variables such as centre.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height, weight and body mass index (BMI).

#### 5.1.2. Additional considerations

Demographic characteristics will also be summarized on Enrolled Set for web public disclosure

Subject disposition will be summarized by group using descriptive statistics:

• Number of subjects screened, randomised, vaccinated and withdrawn including withdrawal reasons in each group and overall will be tabulated.

Vital signs will be summarized by group using descriptive statistics at all timepoint(s) the information is collected on Exposed Set and Per-protocol Set.

Summary of important protocol deviations leading to elimination will be tabulated by group. An individual listing will also be provided.

Summary of medical history will be performed on Exposed Set by Medical Dictionary for Regulatory Activities (MedDRA) and preferred term.

Additional analyses by country and/or by site may be performed if deemed necessary

# 5.2. Immunogenicity

# 5.2.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the Per Protocol set for analysis of immunogenicity. If, in any study group and at any timepoint, the percentage of enrolled or vaccinated subjects with serological results excluded from the Per Protocol set for analysis of immunogenicity is 5% or more, a second analysis based on the Full Analysis Set will be performed to complement the Per Protocol analysis.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled)** |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | <ul> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically pooled.</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI pooled.</li> </ul> |
| | <ul> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> </ul> |
| | The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentrations will be calculated at Screening, Day 8 and Day 31 pooled for all subjects.* |
| | <ul> <li>A further exploratory between-groups analysis will be performed at Day 8 or Day 31 using<br/>an ANCOVA model by including study groups, country, age category, and level of<br/>antibodies at Screening as covariates.</li> </ul> |
| Secondary | (US and ex-US data to be considered pooled, then separately) |
| | For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified): |
| | GMCs/GMTs and their 95% CI will be tabulated and represented graphically by formulation (US and ex-US). |
| | Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI by formulation (US and ex-US). |
| | Antibody titer/concentration will be displayed using reverse cumulative curves by |
| | <ul> <li>formulation (US and ex-US).</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points by formulation (US and ex-US).</li> <li>Booster response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by</li> </ul> |
| | group for each formulation (US and ex-US). |
| | Booster responses to PT, FHA and PRN antigens are defined as: |
| | • For subjects with pre-vaccination antibody concentration below the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the assay cut-offs, |
| | • For subjects with pre-vaccination antibody concentration between the assay cut-offs and below 4 times the assay cut-offs: post-vaccination antibody concentration ≥ 4 times the pre-vaccination antibody concentration, and |

| Endpoint | Statistical Analysis Methods |
|---|---|
| | <ul> <li>For subjects with pre-vaccination antibody concentration ≥ 4 times the assay cut-offs:<br/>post-vaccination antibody concentration ≥ 2 times the pre-vaccination antibody<br/>concentration.</li> </ul> |
| | <ul> <li>The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for each formulation (US and ex-US).</li> </ul> |
| | <ul> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo<br/>in terms of anti-PT, anti-FHA, anti-PRN, anti-D, anti-T will be calculated at Screening<br/>and Day 31 pooled for all subjects and by formulation (US and ex-US).</li> </ul> |
| | <ul> <li>A further exploratory between-groups analysis will be performed at Day 31 using an<br/>ANCOVA model by including study groups, age category, country and level of<br/>antibodies at Screening as covariates.</li> </ul> |
| | <ul> <li>For Boostrix booster response to antigens PT, FHA and PRN, the two-sided<br/>standardized asymptotic 95% CI for the group differences in the percentage of<br/>subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine<br/>group and (minus) the dTpa Placebo vaccine group on Day 31 post vaccination will<br/>be calculated for each formulation.</li> </ul> |
| | <ul> <li>For Boostrix seroprotection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for each formulation.</li> </ul> |
| Will doTertiary | Will be described in a seperate Statistical Analysis . |

<sup>\*</sup>The statistical method will not be applied to primary endpoint. For detailed rationale, refer to Section 8.

#### 5.2.2. Additional considerations

At first analysis at Day 31 and final analysis at Day 181, immunogenicity analysis will be performed on PPS.

#### 5.2.2.1. Between group analysis

This analysis is exploratory. RSVPreF3 IgG antibody concentrations, RSV-A neutralizing antibody titers will applied to following model.

For the analysis of subjects at visit 3 (Day 31), the model will be explored and fitted via the proc glm procedure according to the following code:

```
PROC glm data=sero;
  CLASS group;
  MODEL log_val = baseline group age_cat country_US
country_BE
  Output out= pred;
  LSMEANS group/pdiff cl alpha=0.1;
RUN;
```

<sup>\*\*</sup>pooled group definition is detailed in Table 2

where **log\_val** represents the log-transformed antibody value of the immunogenicity variable at a given post baseline timepoint (Day 31), **baseline** is pre-vaccination logarithm10 transformation of the concentrations/titers, **group** indicates the study group, pooled groups (US and ex-US) will considered in model then separate by formulation. **age\_cat** is indicator variable (0/1) and will be treated as continuous in the model, if the age category at vaccination between 18 - 32 years, otherwise age\_cat equals 1 if age category is between 33 - 45 years at vaccination. **Country\_US** is indicator variable (0/1) and will treated as continuous in the model, if subject from US, then variable will equal to 1, otherwise equals to 0, **Country\_BE** is indicator variable (0/1) and will treated as continuous in model, if subject from BE, then variable equals to 1, otherwise equals to 0, if subject is from Canada, above two indicators equal to 0. The inclusion of age category at vaccination, in the model depends on the availability of the variable and the necessity, therefore, the above SAS code serves as a reference and may be adjusted according to the analysis needs.

GMT/GMC ratios between vaccine groups obtained using above model will be calculated by exponentiating mean difference of logarithm- transformed titres. The 90% CI for GMT/GMC ratio will be obtained by exponential-transformation of the CI for the group least square mean of the log-transformed titres/concentration from the above model.

# 5.2.2.2. Percentage difference between two groups

We will conduct percentage difference of booster responses [Camargo, 1984; Melville -Smith, 1983]. with the two-sided standardized asymptotic 95% CI for dTpa vaccine group when given alone and co-administered with RSVPreF3 by formulation at Day 31.

Percentage difference of protection rate [Vidor, 2008] with the two-sided standardized asymptotic 95% CI for RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group by formulation at Day 31 will be calculated

# 5.3. Analysis of safety and reactogenicity

# 5.3.1. Analysis of safety and reactogenicity planned in the protocol

The following safety analyses will be performed based on the Exposed Set. The following safety analysis will be performed on the pooled data then the US and ex-US separately.

| Endpoint | Statistical Analysis Methods |
|---|---|
| Primary | (US + ex-US data to be pooled) |
| | The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day as well as180-day follow up will be tabulated with exact 95% CI by study group. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits. |
| | The percentage of subjects reporting each individual solicited local AE (any grade, Grade 3 and those resulting in a medically attended visit) and solicited general AE (any grade, Grade 3, any |

209141 (RSV MAT-011) Statistical Analysis Plan

| Endpoint | Statistical Analysis Methods |
|---|---|
| | related, Grade 3 related and those resulting in a medically attended visit) during the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) will be tabulated based on maximum intensity for each group. |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period will be tabulated for each group. Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | The percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e. on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA Preferred Terms and reported during the 30-day follow-up period will be tabulated with exact 95% CI. SAEs will also be described in detail. |
| | The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period and during the 30-day follow-up period will be summarized by each group and pooled. |
| Secondary | (US and ex-US data to be considered pooled, then separately) |
| | The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% CI by study group for each formulation (US and ex-US). The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for AEs resulting in medically attended visits. |
| | The percentage of subjects reporting each individual solicited local AE (any grade, Grade 3 and those resulting in a medically attended visit) and solicited general AE (any grade, Grade 3, any related, Grade 3 related and those resulting in a medically attended visit) during the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) will be tabulated based on maximum intensity for each group for each formulation (US and ex-US). |
| | For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period will be tabulated for each group for each formulation (US and ex-US). Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 or above (> 39.0°C/102.2°F) causally related fever, and fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after each vaccination. |
| | For each formulation (US and ex-US), the percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e. on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be |

| Endpoint | Statistical Analysis Methods |
|---|---|
| | reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. |
| | The percentage of subjects with at least one report of SAE classified by the MedDRA Preferred Terms and reported during the 30-day follow-up period will be tabulated with exact 95% CI for each formulation (US and ex-US), reported during the entire study period (from vaccination up to day 181) will be tabulated with exact 95% CI for each formulation (US and ex-US), pooled formulations and pooled all groups receiving RSVPreF3 will also be described in detail. |
| | The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) from vaccination up to day 181 will be summarized by each group for each formulation (US and ex-US), |
| Tertiary | Will be described in a separate Statistical Analysis Plan |

#### 5.3.2. Additional considerations

# 5.3.2.1. Analysis of solicited events

The analysis of solicited events will be performed on Solicited Safety Set. The intensity of the following solicited events will be assessed as described:

 Table 5
 Intensity scales for solicited symptoms in adults

| | Adults/Child | (≥6 years) |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | collection questionn | contained Clinical Outcome Assessment data naires or indices, which are protected by third is and therefore have been excluded. |
| Redness at injection site Swelling at injection site Temperature* | | |
| Headache | | |
| Fatigue | | |
| Gastrointestinal symptoms<br>(nausea, vomiting, diarrhoea and/or<br>abdominal pain) | | |

The maximum intensity of solicited administration site redness/swelling will be scored at GSK Biological as follows:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Duration in days of solicited local and general adverse events within 7 days after vaccination will be tabulated by study group and overall, and if needed by age group. The derivation rule of duration in days for solicited events is detailed in section 10.1.3.9.

# 5.3.2.2. Analysis of Unsolicited Adverse Events

The analysis of unsolicited events will be performed on Exposed Set.

#### 5.3.2.3. Combined Solicited and Unsolicited Adverse Events

The combined analysis of solicited and unsolicited events will be performed on Exposed Set. A summary of subjects with all combined solicited and unsolicited adverse events will be provided.

Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term code | Corresponding<br>Lower level term<br>decode |
|---|---|---|
| Pain | Injection site pain | 10022086 |
| Redness | Redness at injection site | 10022098 |
| Swelling | Swelling at injection site | 10053425 |
| Fatigue | Fatigue | 10016256 |
| Fever | Fever | 10016558 |
| Headache | Headache | 10019211 |
| Gastrointestinal symptoms <sup>†</sup> | Gastrointestinal disorder | 10017944 |

Please note – to check for AE term in cDISC during dry run

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

#### 5.3.2.4. Other analysis

Other safety analysis will be performed on Exposed Set.

Concomitant medications/products will be coded using the GSKDRUG dictionary. The number and percentage of subjects taking concomitant medications (any medication, any

<sup>†</sup>Gastrointestinal symptoms include nausea, vomiting, diarrhoea and/or abdominal pain.

antipyretic and any antipyretic taken prophylactically, respectively) within 7 days following vaccination, 30 days following vaccination and 6 months following vaccination will be summarized by group. A listing will also be provided.

#### 6. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterise the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for most of these comparisons.

### 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

# 7.1.1. First and final study

Analyses to evaluate objectives and endpoints will be performed in steps.

A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints pertaining to safety and immunogenicity up to Day 31 are available. At this point, the statistician will be unblinded (i.e. individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblinded some specific subjects, the study will be considered as single-blind from this point onwards, with subjects and investigators remaining blinded up to study end. The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

The final end-of-study analysis will be performed when all data for at least primary and secondary endpoints up to study conclusion are available. Individual listings will only be provided at this stage. An integrated clinical study report containing all available data will be written and made available to the investigators.

The final study report will contain at least the final analyses of all primary and secondary endpoints. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These analyses will be documented in annex(es) to the study report and will be made available to the investigators at that time

| Description | Disclosure Purpose<br>(CTRS=public posting, SR=study report,<br>internal) |
|---|---|
| Final Analysis (E1_01) | Public disclosure, Study report |
| First Analysis (E1_02) | Public disclosure |

# 7.2. Statistical considerations for interim analyses

NA

#### 8. CHANGES FROM PLANNED ANALYSES

The calculation of GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentrations will be calculated at Screening, Day 8 and Day 31 pooled for all subjects will remove from analyses plan, since we will report adjusted GMT/GMC ratio and their 90% CI which is generated from ANCOVA model.

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section **** 

#### 9.1. Data derivation

## 9.1.1. Immunogenicity

For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

- For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude subjects with a missing or non-evaluable measurement.
- For the between group assessments, statistical model will be fitted based on the subjects having a result at both the baseline and the considered timepoint.

Following table will demonstrate all antigens will be analysed at considered time point for different treatment groups

| | Immunogenicity<br>Endpoints | Statistical Analysis Methods |
|---|---|---|
| RSVPreF3 | <ul> <li>RSVPreF3 IgG antibody concentration, and</li> <li>Neutralizing antibody titers against RSV-A</li> </ul> | <ul> <li>(US and ex-US data to be considered pooled, then separately)</li> <li>GMCs/GMTs and their 95% CI will be tabulated and represented graphically</li> <li>Geometric mean of ratios of antibody titer/concentrations at each individual post-vaccination time point over pre-vaccination (screening) will be tabulated with 95% CI</li> <li>Antibody titer/concentration will be displayed using reverse cumulative curves pooled.</li> <li>The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points pooled.</li> <li>A further exploratory between-groups of RSVPreF3 dTpa and RSVPreF3 alone in terms of RSV-A Nab titers and RSV IgG antibody concentration, analysis will be performed at Day 31 using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates</li> </ul> |

209141 (RSV MAT-011) Statistical Analysis Plan

| | Immunogenicity<br>Endpoints | Statistical Analysis Methods |
|---|---|---|
| Boostrix<br>(dTpa) | Booster response to PT Booster response to FHA Booster response to PRN | <ul> <li>For the subjects received RSVPreF3 dTpa and subjects received dTpa placebo</li> <li>Booster response rates for PT, FHA and PRN (with exact 95% CI) will be calculated by group for US and ex-US pooled formulation and separately.</li> <li>The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-PT, anti-FHA, anti-PRN will be calculated between Day 31 over Screening for US and ex-US pooled data and separately.</li> <li>A further exploratory between-groups analysis will be performed at Day 31 using an ANCOVA model by including study groups, country, age category, and level of antibodies at Screening as covariates</li> <li>For Boostrix booster response to antigens PT, FHA and PRN, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with a booster response to each antigen in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately</li> </ul> |
| | Anti-D concentration Anti-T concentration | For the subjects received RSVPreF3 dTpa and subjects received dTpa placebo • The percentage of subjects with anti-D antibody concentrations ≥1.0 IU/mL by ELISA and the percentage of subjects with anti-T antibody concentrations ≥1.0 IU/mL by ELISA (with exact 95% CI) will be calculated by group for US and ex-US pooled data and separately • The GMT/GMCs ratio and their 90% CI between RSVPreF3 dTpa and dTpa placebo in terms of anti-D, anti-Twill be calculated at Screening and Day 31 for US and ex-US pooled data and separately. • Protection rate (percentage of subjects with antibody concentrations ≥ 0.1 IU/mL by ELISA) for antigens D and T, the two-sided standardized asymptotic 95% CI for the group differences in the percentage of subjects with antibody concentrations ≥0.1 IU/mL in the RSVPreF3 dTpa vaccine group and (minus) the dTpa Placebo vaccine group at Day 31 post vaccination will be calculated for US and ex-US pooled data and separately. |

# 9.1.1.1. Laboratory assays cut-offs for humoral immunity (Antibody determination)

A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay. The cut-off tests for immunogenicity evaluation will be as per following:

| System | Component | Method | Unit | Cut-off* | ULOQ |
|---|---|---|---|---|---|
| Serum | Respiratory Syncytial Virus A<br>Ab neutralizing | NEU | ED60 and/or IU<br>(international unit) | 18 for ED60<br>TBD for IU | TBD |
| Serum | Respiratory Syncytial Virus<br>PreF3 Ab.IgG concentration | ELI | ELU/mL | 25 | TBD |
| Serum | Bordetella<br>pertussis.Filamentous<br>Hemaglutinin Ab.lgG | ELI | IU/mL | 2.046 | TBD |
| Serum | Bordetella pertussis.Pertactin<br>Ab.lgG | ELI | IU/mL | 2.187 | TBD |
| Serum | Bordetella<br>pertussis.Pertussis Toxin<br>Ab.lgG | ELI | IU/mL | 2.693 | TBD |
| Serum | Corynebacterium<br>diphtheriae.Diphtheria Toxoid<br>Ab.lgG | ELI | IU/mL | 0.057 | TBD |
| Serum | Clostridium tetani.Tetanus<br>Toxoid Ab.lgG | ELI | IU/mL | 0.043 | TBD |

Ab = antibody; ELI = Enzyme-linked immunosorbent assay (ELISA); IgG = immunoglobulin G; RSV = respiratory syncytial virus; ED60 = serum dilution inducing 60% inhibition in plaque forming units; IU/ml = International units/milliliter, IU= International units

Assay cut-off and unit might be subject to change before starting of testing (e.g. in case of requalification, revalidation or standardisation). In this case, this will be documented in the clinical report.

#### 9.2. Statistical Method

NA

#### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section **** (additional study-specific rules).

### 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

### 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

#### 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

# 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

#### 10.1.3.2. Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

#### 10.1.3.3. Height

Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows:

Height in centimeters = Height in inches  $\times 2.54$ 

#### 10.1.3.4. Body mass index (BMI)

BMI will be calculated as follows:

 $BMI = (Weight in kilograms) / (Height in meters)^2$ 

#### **10.1.3.5. Temperature**

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

#### 10.1.3.6. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

## 10.1.3.7. Geometric mean titres (GMTs) and concentrations (GMCs)

Geometric Mean Titre (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Antibody titres or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

#### 10.1.3.8. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.9. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited adverse event period.

# 10.1.3.10. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.11. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a subject following multiple vaccines will be counted as only one occurrence.

# 10.1.4. Display of decimals

#### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group

Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.

Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

#### 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

#### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values are below 10kg where one decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with one decimal.

#### 10.1.4.4. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| <b>GMT or GMC value</b> | Number of decimals to display |
|-------------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

## 10.1.5. Statistical methodology

#### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [, 1934].

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Miettinen and Nurminen [, 1985].

## 10.2. TFL TOC

The Table Figure Listing (TFL) Table Of Content (TOC) which itemizes the planned list of TFL and their associated lay-out is developed as a separate document.

## 11. REFERENCES

Camargo ME, Silveira L, Furuta JA, Oliveira EP, Germek OA. Immunoenzymatic assay of anti-diphtheric toxin antibodies in human serum. *J Clin Microbiol*. 1984 Oct;20(4):772-4.

Christy C, Pichichero ME, Reed GF, Effect of Gender, Race, and Parental Education on Immunogenicity and Reported Reactogenicity of Acellular and Whole-Cell Pertussis Vaccines. Pediatrics (1995), 96(3)

Melville-Smith ME, Seagroatt VA, Watkins JT. A comparison of enzyme-linked immunosorbent assay (ELISA) with the toxin neutralization test in mice as a method for the estimation of tetanus antitoxin in human sera. *J Biol Stand*. 1983 Apr;11(2):137-44.

Vidor E, Plotkin SA. Immunogenicity of a two-component (PT & FHA) acellular pertussis vaccine in various combinations *Hum Vaccin*. 2008 Sep-Oct;4(5):328-40.